CLINICAL TRIAL: NCT03593356
Title: Household Income and Child Development in the First Three Years of Life (Phase 1) Household Income and Child Development in the First Years of Life (Phase 2)
Brief Title: Baby's First Years
Acronym: BFY
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Columbia University (Other); University of Wisconsin, Madison (Other); New York University (Other); University of Maryland (Other); University of Nebraska (Other); University of Minnesota (Other); University of New Orleans (Other); University of Michigan (Other); Duke University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Greg Duncan, Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 20163336; R01HD087384 (NIH); 2R01HD087384 (NIH)
Record Dates: First submitted 2018-05-29; First posted 2018-07-20 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Child Development; Brain Development; Household and Family Processes
Keywords: Poverty; Income; Child Development; Brain Development

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant
Masking Description: Researchers know about amount of cash payment subjects receive at the point of enrollment because they assist subjects with credit card activation and instructions. For follow-up assessments at age 1, 2, 3, 4, 6, 8 interviewers will be blind to the extent possible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monthly cash gift payments of $333 (Experimental): These subjects receive $333 each month for 76 months via debit card.
  Interventions: Behavioral: Monthly cash gift payments of $333
- Monthly cash gift payments of $20 (Active Comparator): These subjects receive $20 each month for 76 months via debit card.
  Interventions: Behavioral: Monthly cash gift payments of $20

INTERVENTIONS:
Behavioral: Monthly cash gift payments of $333 — These subjects receive $333 each month for 76 months via debit card.
  Arms: Monthly cash gift payments of $333
Behavioral: Monthly cash gift payments of $20 — These subjects receive $20 each month for 76 months via debit card.
  Arms: Monthly cash gift payments of $20

SUMMARY:
Recent advances in developmental neuroscience suggest that experiences early in life can have profound and enduring influences on the developing brain. Family economic resources shape the nature of many of these experiences, yet the extent to which they affect children's development is unknown. The project's team of neuroscientists, economists and developmental psychologists is seeking to fill important gaps in scientific knowledge about the role of economic resources in early development by evaluating the first U.S. randomized controlled trial to determine whether unconditional cash gift payments have a causal effect on the cognitive, socio-emotional and brain development of infants and toddlers in low-income U.S. families.

Specifically, 1,000 mothers of infants with incomes below the federal poverty line from four diverse U.S. communities were recruited from post-partum wards and are receiving monthly cash gift payments by debit card for the first 76 months of the child's life. Parents in the experimental group and receiving $333 per month ($3,996 per year), whereas parents in the active comparator group are receiving a nominal monthly payment of $20. In order to understand the impacts of the added income on children's cognitive and behavioral development, the investigators are assessing treatment group differences at ages 4 (this lab assessment was postponed from age 3 to age 4 due to Covid-19), 6, and 8 in lab-administered measures of cognitive, language, and self-regulation development and maternal reports of socio-emotional development. A number of other maternal-reported child outcome measures were gathered at ages 1, 2 and 3. Brain circuitry may be sensitive to the effects of early experience even before early behavioral differences can be detected. In order to understand the impacts of added income on children's brain functioning at age 4, 6, and 8, the investigators will assess, during a lab visit, experimental/active comparator group differences in measures of brain activity (electroencephalography [EEG]). The targeted age for each data collection wave is around the child's birthday, i.e. at 12 months, 24 months, 36 months, 48 months, 72 months, and 96 months.

To understand how family economic behavior, parenting, and parent stress and well-being change in response to income enhancement, the investigators will assess experimental/active comparator differences in family expenditures, food insecurity, housing and neighborhood quality, family routines and time use, parent stress, mental health and cognition, parenting practices, and child care and preschool arrangements. School readiness and outcomes are being assessed at ages 6 and 8. This study will thus provide the first definitive understanding of the extent to which income plays a causal role in determining early child cognitive, socio-emotional and brain development among low-income families.

DETAILED DESCRIPTION:
In the Baby's First Years (BFY) study, one thousand infants born to mothers with incomes falling below the federal poverty threshold in four metropolitan areas in the United States were assigned at random within each of the metropolitan areas to one of two cash gift conditions. The sites are: New York City, the greater New Orleans metropolitan area, the greater Omaha metropolitan area, and the Twin Cities. IRB and recruiting issues led to a distribution of the 1,000 mothers across sites of 121 in one site (the Twin Cities), 295 in two of the other sites (New Orleans and Omaha) and 289 in New York. (The investigators have also randomly sampled 80 of the participating families in the Twin Cities and New Orleans to participate in an in-depth qualitative study, but do not elaborate on those plans in this document.) Mothers were recruited in postpartum wards of the 12 participating hospitals shortly after giving birth and, after consenting, were administered a 30-minute baseline interview. They then were asked to agree to receive the cash gifts. The "high-cash gift" treatment group mothers (40% of all mothers) are receiving unconditioned cash payments of $333 per month ($4,000 per year) via debit card for 76 months. Mothers in the "low-cash gift" comparator group (60% of all mothers) are receiving a nominal payment - $20 per month, delivered in the same way and also for 76 months. The 40/60 randomization assignment is stratified by site, but not by hospitals, within each of the four sites. The investigators have worked with state and local officials to ensure that, to the extent feasible, the cash gifts payments are not considered countable income for the purposes of determining benefit levels from social assistance programs.

BFY was originally formulated to study the effects of monthly unconditional cash transfers on child development for the first three years of life, with the cash gifts set to be distributed for 40 months (3 years, 4 months). In response to the COVID-19 pandemic and the need to postpone in-person research activities, the cash transfers were extended for an additional year, through 52 months (4 years, 4 months), enabling us to postpone in-person direct child assessments to age 4. The investigators successfully arranged funding to extend the cash gifts for a total of 76 months - the approximate boundary between early and middle childhood - and informed the study participants in August 2022 about the additional 2-year extension of cash transfer.

The targeted age for each data collection wave is around the child's birthday, i.e. at 12 months, 24 months, 36 months, 48 months, 72 months, and 96 months. Interviews conducted at child ages 1, 2 and 3 provided information about family functioning as well as several maternal reports of developmentally-appropriate measures of children's cognitive and behavioral development. At ages 4, 6 and 8 measures of cognitive, language, and self-regulation development were or will be administered in university labs, while socio-emotional development is assessed via maternal report. EEG-based measures of brain activity were assessed in the home at age 1 and in labs at ages 4, 6 and 8. At age 6 and 8 the investigators will collect school behavior and engagement data.

Conditional on participants' consent and our success in securing agreements with state and county agencies, the investigators are also collecting state and local administrative data regarding parental employment, utilization of public benefits such as Medicaid and Supplemental Nutrition Assistance Programs (SNAP), and any involvement in child protective services.

The family process measures that the investigators will gather are based on two theories of change surrounding the income supplements: that increased investment and reduced stress will facilitate children's healthy development. The investigators are obtaining measures of both of these pathways annually. Investment pathway: Additional resources enable parents to buy goods and services for their families and children that support cognitive development. These include higher quality housing, nutrition and non-parental child care; more cognitively stimulating home environments and learning opportunities outside of the home; and, by reducing or restructuring work hours, more parental time spent with children. Stress pathway: A second pathway is that additional economic resources may reduce parents' own stress and improve their mental health. This may allow parents to devote more positive attention to their children, thus providing a more predictable family life, less conflicted relationships, and warmer and more responsive interactions.

The compensation difference between families in the high and low cash gift groups will boost family incomes by $3,760 per year, an amount shown in the economics and developmental psychology literatures to be associated with socially significant and policy relevant improvements in children's school achievement. After accounting for likely attrition, a total sample size of 800 at age 4, 6 and 8 years, divided 40/60 between high and low payment groups, provides sufficient statistical power to detect meaningful (roughly .20 SD) differences in cognitive, emotional and brain functioning, and key dimensions of family context.

Measures and preregistered hypotheses about child- and family-based measures at all data collection waves are shown in the two tables in the Statistical Analysis Plan in "Other Documents" below; child-focused preregistered hypotheses are presented in Appendix Table 9 and maternal and family focused preregistered hypotheses are presented in Appendix Table 10. The investigators will update this registry with Age 8 measures and preregistered hypotheses before data collection begins in July 2026. The lab-based assessments at child ages 6 and 8 are part of Phase 2 of the project. The Phase 1 analysis plan covers ages 1-4.

ELIGIBILITY:
Inclusion Criteria:

1. mother 18 years or older;
2. household income below the federal poverty threshold in the calendar year prior to the interview, counting the newborn;
3. infant admitted to the newborn nursery and not requiring admittance to the intensive care unit;
4. residence in the state of recruitment;
5. mother not "highly likely" to move to a different state or country in the next 12 months;
6. infant to be discharged in the custody of the mother;
7. English or Spanish speaking (necessary for administration of instruments used to measure some of the child outcomes);
8. singleton birth

Exclusion Criteria:

Mothers will not be eligible unless all of the above eight criteria are met.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligibility: Mothers who just gave birth
Enrollment: 1000 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-08-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Greg Duncan, PhD, Study Director — University of California, Irvine
Locations (1):
- 12 hospitals in the following four metropolitan areas: New York, Omaha, New Orleans, and Twin Cities, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Troller-Renfree SV, Morales S, Leach SC, Bowers ME, Debnath R, Fifer WP, Fox NA, Noble KG. Feasibility of assessing brain activity using mobile, in-home collection of electroencephalography: methods and analysis. Dev Psychobiol. 2021 Sep;63(6):e22128. doi: 10.1002/dev.22128. Epub 2021 Jun 4. PMID 34087950
- [Result] Troller-Renfree SV, Sperber JF, Hart ER, Costanzo MA, Gennetian LA, Meyer JS, Fox NA, Noble KG. Associations between maternal stress and infant resting brain activity among families residing in poverty in the U.S. Biol Psychol. 2023 Nov;184:108683. doi: 10.1016/j.biopsycho.2023.108683. Epub 2023 Sep 15. PMID 37716521
- [Result] Costanzo MA, Magnuson KA, Gennetian LA, Halpern-Meekin S, Noble KG, Yoshikawa H. Contraception use and satisfaction among mothers with low income: Evidence from the Baby's First Years study. Contraception. 2024 Jan;129:110297. doi: 10.1016/j.contraception.2023.110297. Epub 2023 Oct 6. PMID 37806470
- [Result] Sperber JF, Gennetian LA, Hart ER, Kunin-Batson A, Magnuson K, Duncan GJ, Yoshikawa H, Fox NA, Halpern-Meekin S, Noble KG. Unconditional Cash Transfers and Maternal Assessments of Children's Health, Nutrition, and Sleep: A Randomized Clinical Trial. JAMA Netw Open. 2023 Sep 5;6(9):e2335237. doi: 10.1001/jamanetworkopen.2023.35237. PMID 37773497
- [Result] Premo EM, Magnuson KA, Lorenzo NE, Fox NA, Noble KG. Mental health and sleep quality of low-income mothers of one-year-olds during the COVID-19 pandemic. Infant Ment Health J. 2023 Jul;44(4):572-586. doi: 10.1002/imhj.22074. PMID 37439103
- [Result] Troller-Renfree SV, Hart ER, Sperber JF, Fox NA, Noble KG. Associations among stress and language and socioemotional development in a low-income sample. Dev Psychopathol. 2022 May;34(2):597-605. doi: 10.1017/S0954579421001759. Epub 2022 Mar 8. PMID 35256040
- [Result] Collins JM, Halpern-Meekin S, Harvey M, Hoiting J. "I Don't Like All Those Fees" Pragmatism About Financial Services Among Low-Income Parents. J Fam Econ Issues. 2022 Nov 5:1-14. doi: 10.1007/s10834-022-09873-w. Online ahead of print. PMID 36373018
- [Result] Yoo PY, Duncan GJ, Magnuson K, Fox NA, Yoshikawa H, Halpern-Meekin S, Noble KG. Unconditional cash transfers and maternal substance use: findings from a randomized control trial of low-income mothers with infants in the U.S. BMC Public Health. 2022 May 5;22(1):897. doi: 10.1186/s12889-022-12989-1. PMID 35513842
- [Result] Noble KG, Magnuson K, Gennetian LA, Duncan GJ, Yoshikawa H, Fox NA, Halpern-Meekin S. Baby's First Years: Design of a Randomized Controlled Trial of Poverty Reduction in the United States. Pediatrics. 2021 Oct;148(4):e2020049702. doi: 10.1542/peds.2020-049702. Epub 2021 Sep 2. PMID 34475270
- [Result] Troller-Renfree SV, Costanzo MA, Duncan GJ, Magnuson K, Gennetian LA, Yoshikawa H, Halpern-Meekin S, Fox NA, Noble KG. The impact of a poverty reduction intervention on infant brain activity. Proc Natl Acad Sci U S A. 2022 Feb 1;119(5):e2115649119. doi: 10.1073/pnas.2115649119. PMID 35074878
- [Result] Adams EJ, Scott ME, Amarante M, Ramirez CA, Rowley SJ, Noble KG, Troller-Renfree SV. Fostering inclusion in EEG measures of pediatric brain activity. NPJ Sci Learn. 2024 Apr 2;9(1):27. doi: 10.1038/s41539-024-00240-y. PMID 38565857
- [Result] Collins JM, Halpern-Meekin S, Harvey M, Hoiting J. "If I don't have credit, I don't have anything": Perspectives on the credit scoring system among mothers with low incomes. J Consum Aff. 2023 Winter;57(4):1605-1622. doi: 10.1111/joca.12561. Epub 2023 Sep 30. PMID 38214004
- [Result] Barnes C, Halpern-Meekin S, Hoiting J. "I Used to Get WIC... But Then I Stopped": How WIC Participants Perceive the Value and Burdens of Maintaining Benefits. RSF. 2023 Sep;9(5):32-55. doi: 10.7758/rsf.2023.9.5.02. PMID 38486832
- [Result] Gennetian LA, Duncan G, Fox NA, Halpern-Meekin S, Magnuson K, Noble KG, Yoshikawa H. Unconditional Cash and Family Investments in Infants: Evidence from a Large-Scale Cash Transfer Experiment in the U.S. Res Sq [Preprint]. 2023 Feb 7:rs.3.rs-2507540. doi: 10.21203/rs.3.rs-2507540/v1. PMID 36798246
- [Result] Gennetian LA, Duncan GJ, Fox NA, Halpern-Meekin S, Magnuson K, Noble KG, Yoshikawa H. Effects of a monthly unconditional cash transfer starting at birth on family investments among US families with low income. Nat Hum Behav. 2024 Aug;8(8):1514-1529. doi: 10.1038/s41562-024-01915-7. Epub 2024 Jun 21. PMID 38907028
- [Result] Halpern-Meekin S, Gennetian LA, Hoiting J, Stilwell L, Meyer L. Monthly unconditional income supplements starting at birth: Experiences among mothers of young children with low incomes in the U.S. J Policy Anal Manage. 2024 Summer;43(3):871-898. doi: 10.1002/pam.22571. Epub 2024 Mar 2. PMID 39035030
- [Result] Egan-Dailey S, Gennetian LA, Magnuson K, Duncan GJ, Yoshikawa H, Fox NA, Noble KG. Child-directed speech in a large sample of U.S. mothers with low income. Child Dev. 2024 Nov-Dec;95(6):2045-2061. doi: 10.1111/cdev.14139. Epub 2024 Jul 29. PMID 39073390
- [Result] Das A, Osypuk TL, Yoo PY, Magnuson K, Gennetian LA, Noble KG, Bruckner TA. Poverty reduction and childhood opportunity moves: A randomized trial of cash transfers to low-income U.S. families with infants. Health Place. 2024 Sep;89:103320. doi: 10.1016/j.healthplace.2024.103320. Epub 2024 Aug 2. PMID 39096582
- [Result] Hart ER, Gennetian LA, Sperber JF, Penalva R, Magnuson K, Duncan GJ, Halpern-Meekin S, Yoshikawa H, Fox NA, Noble KG. The effect of unconditional cash transfers on maternal assessments of children's early language and socioemotional development: Experimental evidence from U.S. families residing in poverty. Dev Psychol. 2024 Dec;60(12):2290-2305. doi: 10.1037/dev0001824. Epub 2024 Aug 22. PMID 39172428
- [Result] Stilwell L, Morales-Gracia M, Magnuson K, Gennetian LA, Sauval M, Fox NA, Halpern-Meekin S, Yoshikawa H, Noble KG. Unconditional Cash and Breastfeeding, Child Care, and Maternal Employment among Families with Young Children Residing in Poverty. Soc Serv Rev. 2024 Jun;98(2):260-292. doi: 10.1086/729364. Epub 2024 May 22. PMID 39148861
- [Derived] Duncan GJ, Magnuson K, Kunin-Batson AS, Yoshikawa H, Fox NA, Halpern-Meekin S, Ainsworth NJ, Black SR, Nelson JM, Nelson TD, Georgieff MK, Karhson D, Gennetian LA, Noble KG. Cash Transfers and Their Effect on Maternal and Young Children's Health: A Randomized Clinical Trial. JAMA Pediatr. 2025 Aug 1;179(8):867-875. doi: 10.1001/jamapediatrics.2025.1612. PMID 40522644
- [Derived] Sperber JF, Gennetian LA, Hart ER, Kunin-Batson A, Magnuson K, Duncan GJ, Yoshikawa H, Fox NA, Halpern-Meekin S, Noble KG. The Effect of a U.S. Poverty Reduction Intervention on Maternal Assessments of Young Children's Health, Nutrition, and Sleep: A Randomized Control Trial. medRxiv [Preprint]. 2023 May 26:2023.05.25.23290530. doi: 10.1101/2023.05.25.23290530. PMID 37292982
- See also: This website is for Study Participants for general study information and contact information. — http://www.4mybabycard.com
- See also: Study Research Website — http://www.babysfirstyears.com

RESULTS

PARTICIPANT FLOW:
Period: Age 1 Wave
Arm/Group | Monthly Cash Gift Payments of $333 | Monthly Cash Gift Payments of $20
Started | 400 | 600
Completed | 383 | 548
Not Completed | 17 | 52
Period: Age 2 Wave
Arm/Group | Monthly Cash Gift Payments of $333 | Monthly Cash Gift Payments of $20
Started | 397 | 599
Completed | 377 | 545
Not Completed | 20 | 54
Period: Age 3 Wave
Arm/Group | Monthly Cash Gift Payments of $333 | Monthly Cash Gift Payments of $20
Started | 397 | 598
Completed | 380 | 542
Not Completed | 17 | 56
Period: Age 4 Wave
Arm/Group | Monthly Cash Gift Payments of $333 | Monthly Cash Gift Payments of $20
Started | 395 | 589
Completed | 375 | 517
Not Completed | 20 | 72

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Monthly Cash Gift Payments of $333 | Monthly Cash Gift Payments of $20 | Total
Number analyzed (Participants) | 400 | 600 | 1000
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 400 | 600 | 1000
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.38 (5.86) | 26.80 (5.82) | 27.03 (5.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 400 | 600 | 1000
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non-Hispanic | 34 | 67 | 101
  Black, non-Hispanic | 177 | 237 | 414
  Multiple races, non-Hispanic | 12 | 24 | 36
  Other race, non-Hispanic or unknown | 11 | 29 | 40
  Hispanic | 166 | 243 | 409
Region of Enrollment [Number; unit: participants]
  United States | 400 | 600 | 1000

OUTCOME MEASURES:

1. Primary Outcome: Child Language Development: Vocabulary
Description: Measured by Receptive One Word Picture Vocabulary Test (ROWPVT). We analyze conceptual vocabulary scores.
  Minimum raw value: 0; Maximum raw value: 111. Higher score indicates a better outcome.
  References:
  Martin, N. A., & Brownell, R. (2011). ROWPVT-4: Receptive One-Word Picture Vocabulary Test.
Time Frame: Age 48 months
Population: An additional 31 participants attempted this assessment but were excluded from analysis for the following reasons: child's behavior or responses did not yield a valid score (n=25); technical error (n=4); experimenter error (n=1); primary language neither English nor Spanish (n=1).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Monthly Cash Gift Payments of $333 | Monthly Cash Gift Payments of $20
Number analyzed (Participants) | 296 | 404
score on a scale | 39.20 (15.52) | 41.00 (16.20)
Statistical Analysis 1: Comparison: Monthly Cash Gift Payments of $333 vs Monthly Cash Gift Payments of $20; Test type: Superiority; p = 0.717, Regression, Linear — We use OLS regression with site fixed effects and baseline covariates. We report unadjusted p-values; Slope = -0.427, Standard Error of Mean 1.179 — Positive (negative) estimates indicate the high cash gift group had a higher (lower) mean than the low cash gift group. Our measure of dispersion of parameter estimates is the standard error of estimate as described in our analysis plan

2. Primary Outcome: Child Language Development: Vocabulary
Description: Expressive One-Word Picture Vocabulary (EOWPVT) monolingual and bilingual version. Score range monolingual version: 0-185, bilingual version: 0-180; higher scores indicate better performance. Because the two versions of the test are not co-normed, the primary outcome will be a derived "conceptual score" or sum of the raw scores on all individual items that appear on both versions of the test. Expect higher scores in high- than low-cash gift group.
  Reference:
  Martin, N., & Brownell, R. (2011). Expressive one-word picture vocabulary test (4th ed.). Novato: Academic Therapy Publications.
Time Frame: Age 6
Reporting Status: Not Posted, anticipated posting 2026-08

3. Primary Outcome: Child Language Development: Vocabulary
Description: Expressive One-Word Picture Vocabulary (EOWPVT) monolingual and bilingual version. Score range monolingual version: 0-185, bilingual version: 0-180; higher scores indicate better performance. Because the two versions of the test are not co-normed, the primary outcome will be a derived "conceptual score" or sum of the raw scores on all individual items that appear on both versions of the test. Expect higher scores in high- than low-cash gift group.
  Reference:
  Martin, N., & Brownell, R. (2011). Expressive one-word picture vocabulary test (4th ed.). Novato: Academic Therapy Publications.
  If reporting a score on a scale, please include the unabbreviated scale title, the minimum and maximum values, and whether higher scores mean a better or worse outcome.
Time Frame: Age 8
Reporting Status: Not Posted, anticipated posting 2028-08

4. Primary Outcome: Child Language Development: Maternal Concern for Language Delay
Description: Measured by the sum of the two questions listed below included in the Parents' Evaluation of Developmental Status (PEDS):
  1. Do you have any concerns about how your child talks and makes speech sounds? (0: No; 1: Yes or a little)
  2. Do you have any concerns about how your child understands what you say? (0: No; 1: Yes or a little)".
  Minimum score: 0; Maximum score: 2. Higher score indicates worse outcome.
  We will estimate the statistical significance of the entire family of related measures in the Child Language Development outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Glascoe FP. Parents' Evaluations of Developmental Status: A Method for Detecting and Addressing Developmental and Behavioral Problems in Children. Nashville, TN: Ellsworth & Vandermeer Press, 1997.
Time Frame: Age 36 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Monthly Cash Gift Payments of $333 | Monthly Cash Gift Payments of $20
Number analyzed (Participants) | 377 | 542
units on a scale | 0.36 (0.63) | 0.38 (0.65)
Statistical Analysis 1: Comparison: Monthly Cash Gift Payments of $333 vs Monthly Cash Gift Payments of $20; Test type: Superiority; p = 0.784, Regression, Linear — We reported the Westfall-Young adjusted p-value, using OLS regression with site fixed effects and baseline covariates. The unadjusted p-value was 0.789; Slope = -0.012, Standard Error of Mean 0.043 — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: Child Executive Function & Behavioral Regulation: Executive Function
Description: Executive Function measured by Minnesota Executive Function Scale. We analyze standard scores.
  Minimum score: 60; Maximum score: 140. Higher score indicates a better outcome.
  Reference:
  Carlson, S.M. (2017). Minnesota Executive Function Scale: Technical report.
  Carlson, S. M., & Zelazo, P. D. (2014). Minnesota Executive Function Scale: Test Manual. St. Paul, MN: Reflection Sciences, Inc.
Time Frame: Age 48 months
Population: An additional 31 participants attempted this assessment but were excluded from analysis for the following reasons: child unable/unwilling to complete assessment (n=24); experimenter error (n=4); technical error (n=3).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Monthly Cash Gift Payments of $333 | Monthly Cash Gift Payments of $20
Number analyzed (Participants) | 334 | 449
score on a scale | 94.55 (10.60) | 93.75 (10.48)
Statistical Analysis 1: Comparison: Monthly Cash Gift Payments of $333 vs Monthly Cash Gift Payments of $20; Test type: Superiority; p = 0.474, Regression, Linear — We use OLS regression with site fixed effects and baseline covariates. We report unadjusted p-values; Slope = 0.578, Standard Error of Mean 0.807 — [estimate comment as in outcome 1, analysis 1]

6. Primary Outcome: Child Executive Function & Behavioral Regulation: Executive Function
Description: Measured by the Minnesota Executive Function Scale (MEFS); score range: 0-100; higher scores indicate better performance. Expect higher scores in high- than low-cash gift group.
  Reference:
  Carlson, S.M. (2017). Minnesota Executive Function Scale: Technical report. Carlson, S. M., & Zelazo, P. D. (2014). Minnesota Executive Function Scale: Test Manual. St. Paul, MN: Reflection Sciences, Inc.
Time Frame: Age 6
Reporting Status: Not Posted, anticipated posting 2026-08

7. Primary Outcome: Child Executive Function & Behavioral Regulation: Executive Function
Description: as for outcome 6
Time Frame: Age 8
Reporting Status: Not Posted, anticipated posting 2028-08

8. Primary Outcome: Child Executive Function & Behavioral Regulation: Inhibitory Control and Attention
Description: Measured by the NIH Toolbox Flanker Inhibitory Control and Attention task. Score range: 0-30; higher scores indicate better performance.Expect higher scores in high- than low-cash gift group.
  Reference:
  National Institutes of Health and Northwestern University (2006-2023). NIH Toolbox® for Assessment of Neurological and Behavioral Function Administrator's Manual. NIHToolbox.org.
  Gershon, R. C., Wagster, M. V., Hendrie, H. C., Fox, N. A., Cook, K. F., & Nowinski, C. J. (2013). NIH Toolbox for assessment of neurological and behavioral function. Neurology, 80(11 Suppl 3), S2-S6. https://doi.org/10.1212/WNL.0b013e3182872e5f Weintraub S, Bauer PJ, Zelazo PD, Wallner-Allen K, Dikmen SS, Heaton RK, Tulsky DS, Slotkin J, Blitz DL, Carlozzi NE, Havlik RJ, Beaumont JL, Mungas D, Manly JJ, Borosh BG, Nowinski CJ, Gershon RC. I. NIH Toolbox Cognition Battery (CB): introduction and pediatric data. Monogr Soc Res Child Dev. 2013 Aug;78(4):1-15. doi: 10.1111/mono.12031. PMID: 23952199
Time Frame: Age 6
Reporting Status: Not Posted, anticipated posting 2026-08

9. Primary Outcome: Child Executive Function & Behavioral Regulation: Inhibitory Control and Attention
Description: as for outcome 8
Time Frame: Age 8
Reporting Status: Not Posted, anticipated posting 2028-08

10. Primary Outcome: Child Executive Function & Behavioral Regulation: Working Memory
Description: Measured by the Wechsler Preschool and Primary Scale of Intelligence (WPPSI) picture memory subtest. Picture Memory score range: 0-35, higher scores indicate better performance. Expect higher scores in high- than low-cash gift group.We pre-register three scores (MEFS, Flanker, Picture Memory),with a plan to do a confirmatory factor analysis and pre-register the impact on the common factor.
  Reference:
  Wechsler, D. (2012). Wechsler Preschool and Primary Scale of Intelligence Fourth Edition (WPPSI-IV). San Antonio, TX: The Psychological Corporation.
Time Frame: Age 6
Reporting Status: Not Posted, anticipated posting 2026-08

11. Primary Outcome: Child Executive Function & Behavioral Regulation: Working Memory
Description: Measured by Wechsler Intelligence Scale for Children: 5th Edition (WISC-V) subtest Digit Span. Score Range 0-54. Higher scores indicate better performance. We will pre-register three scores (MEFS, Flanker, Digit Span),with a plan to do a confirmatory factor analysis and pre-register the impact on the common factor. Expect higher scores in high- than low-cash gift group.
  Reference:
  Wechsler, D. (2014). Wechsler Intelligence Scale for Children-Fifth Edition (WISC-V). Bloomington, MN: Pearson.
Time Frame: Age 8
Reporting Status: Not Posted, anticipated posting 2028-08

12. Primary Outcome: Child Socio-Emotional Processing: Behavior/Problems
Description: Behavior/Problems measured by Child Behavior Checklist (CBCL).
  Minimum score: 0; Maximum score: 82. Higher score indicates a better outcome.
  We will estimate the statistical significance of the entire family of related measures in the Child Socio-Emotional Processing outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Achenbach, T. M., & Ruffle, T. M. (2000). The Child Behavior Checklist and related forms for assessing behavioral/emotional problems and competencies. Pediatrics in review, 21(8), 265-271.
Time Frame: Age 36 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Monthly Cash Gift Payments of $333 | Monthly Cash Gift Payments of $20
Number analyzed (Participants) | 378 | 542
units on a scale | 18.42 (13.00) | 18.51 (13.26)
Statistical Analysis 1: Comparison: Monthly Cash Gift Payments of $333 vs Monthly Cash Gift Payments of $20; Test type: Superiority; p = 0.871, Regression, Linear — We reported the Westfall-Young adjusted p-value, using OLS regression with site fixed effects and baseline covariates. The unadjusted p-value was 0.791; Slope = 0.234, Standard Error of Mean 0.882 — [estimate comment as in outcome 1, analysis 1]

13. Primary Outcome: Child Socio-Emotional Processing: Maternal Concern for Behavioral and Social-Emotional Problems
Description: Measured by the sum of the two questions listed below, which are part of the Parents' Evaluation of Developmental Status (PEDS):
  1. Do you have any concerns about how your child behaves? (0: No; 1: Yes or a little)
  2. Do you have any concerns about how your child gets along with others? (0: No; 1: Yes or a little).
  Minimum score: 0; Maximum score: 2. Higher score indicates worse outcome.
  We will estimate the statistical significance of the entire family of related measures in the Child Socio-Emotional Processing outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Glascoe FP. Parents' Evaluations of Developmental Status: A Method for Detecting and Addressing Developmental and Behavioral Problems in Children. Nashville, TN: Ellsworth & Vandermeer Press, 1997.
Time Frame: Age 36 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Monthly Cash Gift Payments of $333 | Monthly Cash Gift Payments of $20
Number analyzed (Participants) | 378 | 542
units on a scale | 0.41 (0.69) | 0.39 (0.67)
Statistical Analysis 1: Comparison: Monthly Cash Gift Payments of $333 vs Monthly Cash Gift Payments of $20; Test type: Superiority; p = 0.871, Regression, Linear — We reported the Westfall-Young adjusted p-value, using OLS regression with site fixed effects and baseline covariates. The unadjusted p-value was 0.646; Slope = 0.021, Standard Error of Mean 0.046 — [estimate comment as in outcome 1, analysis 1]

14. Primary Outcome: Child Socio-Emotional Processing: Behavior/Problems
Description: Behavior/Problems measured by Child Behavior Checklist (CBCL). We analyze a preregistered index (sum of raw scores on 4 subscales: Anxiety/Depression, Aggressive Behavior, Attention Problems, and Emotionally Reactive).
  Minimum score: 0; Maximum score: 82. Higher score indicates a better outcome.
  Reference:
  Achenbach, T. M., & Ruffle, T. M. (2000). The Child Behavior Checklist and related forms for assessing behavioral/emotional problems and competencies. Pediatrics in review, 21(8), 265-271.
Time Frame: Age 48 months
Population: One additional participant attempted this assessment but was excluded because of missing data on more than 80% of items.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Monthly Cash Gift Payments of $333 | Monthly Cash Gift Payments of $20
Number analyzed (Participants) | 369 | 513
score on a scale | 22.39 (12.50) | 22.18 (12.93)
Statistical Analysis 1: Comparison: Monthly Cash Gift Payments of $333 vs Monthly Cash Gift Payments of $20; Test type: Superiority; p = 0.872, Regression, Linear — We use OLS regression with site fixed effects and baseline covariates. We report unadjusted p-values; Slope = 0.139, Standard Error of Mean 0.860 — [estimate comment as in outcome 1, analysis 1]

15. Primary Outcome: Child Socio-Emotional Processing: Behavior/Problems
Description: Measured by the Brief Problem Monitor (BPM), assesses attentional, behavioral, and internalizing problems in children. 19 questions and answer choices. Score range: 0-38; higher scores indicate more behavioral problems. Expect lower scores in high- than low-cash gift group.
  Reference:
  Achenbach, T. M., McConaughy, S. H., Ivanova, M. Y., & Rescorla, L. A. (2011). Manual for the ASEBA Brief Problem Monitor (BPM). Burlington, VT: University of Vermont, Research Center for Children, Youth, & Families.: ASEBA.
Time Frame: Age 6
Reporting Status: Not Posted, anticipated posting 2026-08

16. Primary Outcome: Child Socio-Emotional Processing: Behavior/Problems
Description: as for outcome 15
Time Frame: Age 8
Reporting Status: Not Posted, anticipated posting 2028-08

17. Primary Outcome: Child Brain Function: Resting Brain Function
Description: Measured by high-density in-lab electroencephalography (EEG).
  Because of limitations in power expected with multiple testing adjustments, we are preregistering a single composite of mid-to-high-frequency whole-brain power summing across alpha, beta, and gamma bands, from 7 to 45 Hz. The composite will reflect the sum of power values (μV2) for each 1-Hz frequency bin between 7 and 45 Hz. Please see statistical analysis plan for more details.
  References:
  Tomalski, P., et al. (2013); Otero, G. A., et. al (2003); Marshall, P. J., et.al. (2004)
  Troller-Renfree, S. V., et. al. (2022). The impact of a poverty reduction intervention on infant brain activity. Proceedings of the National Academy of Sciences, 119(5).
Time Frame: Age 48 months
Population: An additional 187 participants were excluded for the following reasons: mother did not consent to EEG collection (n=70), child or parent refused to participate after consenting (n=86), technical problems/experimenter error or ill-fitting cap (n=13), visit ended before EEG collection (n=4), a developmental condition prohibiting collection (n=1), poor data quality (n=4), not enough usable data (n=9).
Measure: Mean (Standard Deviation); unit: μV^2
Arm/Group | Monthly Cash Gift Payments of $333 | Monthly Cash Gift Payments of $20
Number analyzed (Participants) | 278 | 359
μV^2 | 3.05 (1.35) | 2.92 (1.37)
Statistical Analysis 1: Comparison: Monthly Cash Gift Payments of $333 vs Monthly Cash Gift Payments of $20; Test type: Superiority; p = 0.184, Regression, Linear — We use OLS regression with site fixed effects and baseline covariates. We report unadjusted p-values; Slope = 0.133, Standard Error of Mean 0.100 — [estimate comment as in outcome 1, analysis 1]

18. Primary Outcome: Child Brain Function: Resting Brain Function
Description: Measured by high-density in-lab electroencephalography (EEG). Ages 6 and 8 Primary hypothesis: Because of limitations in power expected with multiple testing adjustments, we are preregistering a single composite index of mid-to-high-frequency whole-brain power summed across alpha, beta, and gamma bands (defined as between 7 and 45 Hz). This frequency composite index sums absolute power (μV2) across all single-Hz intervals in the Alpha, Beta, and Gamma bands (7-45 Hz). We hypothesize that, in the eyes-closed condition, the high-cash gift group will show more power in this composite relative to the low-cash gift group. One-tailed t-tests will be used to test this directional hypothesis. See the Statistical Analysis Plan (Phase 2) for additional details and references.
Time Frame: Age 6
Reporting Status: Not Posted, anticipated posting 2026-08

19. Primary Outcome: Child Brain Function: Resting Brain Function
Description: as for outcome 18
Time Frame: Age 8
Reporting Status: Not Posted, anticipated posting 2028-08

20. Primary Outcome: Child Health, Sleep
Description: Measured by an adapted Short Form of Patient-Reported Outcomes Measurement Information System (PROMIS™).
  Minimum score: 3; Maximum score: 15. Higher score indicates a better outcome.
  Reference:
  Yu, L., Buysse, D. J., Germain, A., Moul, D. E., Stover, A., Dodds, N. E., ... & Pilkonis, P. A. (2012). Development of short forms from the PROMIS™ sleep disturbance and sleep-related impairment item banks. Behavioral sleep medicine, 10(1), 6-24.
Time Frame: Age 36 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Monthly Cash Gift Payments of $333 | Monthly Cash Gift Payments of $20
Number analyzed (Participants) | 377 | 542
units on a scale | 5.10 (2.50) | 5.04 (2.61)
Statistical Analysis 1: Comparison: Monthly Cash Gift Payments of $333 vs Monthly Cash Gift Payments of $20; Test type: Superiority; p = 0.415, Regression, Linear — We reported the Westfall-Young adjusted p-value, using OLS regression with site fixed effects and baseline covariates. The unadjusted p-value was 0.427; Slope = 0.138, Standard Error of Mean 0.173 — [estimate comment as in outcome 1, analysis 1]

21. Primary Outcome: Child Health, Overall Health, Medical Care, Diagnosis of Condition or Disability
Description: Measured by an index of six items (see Appendix Table 7 in "Analysis Plan and Measures" document for items).
  Minimum score: 3; Maximum score: 14. Higher score indicates a worse outcome.
  Reference:
  Halim, M. L., Yoshikawa, H., & Amodio, D. M. (2013). Cross-generational effects of discrimination among immigrant mothers: Perceived discrimination predicts child's healthcare visits for illness. Health Psychology, 32(2), 203.
Time Frame: Age 36 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Monthly Cash Gift Payments of $333 | Monthly Cash Gift Payments of $20
Number analyzed (Participants) | 378 | 542
units on a scale | 4.92 (1.96) | 4.91 (2.12)
Statistical Analysis 1: Comparison: Monthly Cash Gift Payments of $333 vs Monthly Cash Gift Payments of $20; Test type: Superiority; p = 0.567, Regression, Linear — We reported the Westfall-Young adjusted p-value, using OLS regression with site fixed effects and baseline covariates. The unadjusted p-value was 0.541; Slope = 0.086, Standard Error of Mean 0.140 — [estimate comment as in outcome 1, analysis 1]

22. Primary Outcome: Child Academic Achievement: Reading
Description: Woodcock Johnson IV Test of Achievement: Letter-Word ID. Score range: 0-78; higher scores indicate better performance. Expect higher scores in high- than low-cash gift group.
  Reference:
  McGrew, K. S., & Woodcock, R. W. (2018). Woodcock-Johnson IV Tests of Achievement. Rolling Meadows, IL: Riverside Publishing.
Time Frame: Age 6
Reporting Status: Not Posted, anticipated posting 2026-08

23. Primary Outcome: Child Academic Achievement: Reading
Description: as for outcome 22
Time Frame: Age 8
Reporting Status: Not Posted, anticipated posting 2028-08

24. Primary Outcome: Child Academic Achievement: Reading Comprehension
Description: Woodcock Johnson IV Test of Achievement: Passage Comprehension. Score range: 0-52. Expect higher scores in high- than low-cash gift group.
  Reference:
  McGrew, K. S., & Woodcock, R. W. (2018). Woodcock-Johnson IV Tests of Achievement. Rolling Meadows, IL: Riverside Publishing.
Time Frame: Age 8
Reporting Status: Not Posted, anticipated posting 2028-08

25. Primary Outcome: Child Academic Achievement: Math
Description: as for outcome 22
Time Frame: Age 6
Reporting Status: Not Posted, anticipated posting 2026-08

26. Primary Outcome: Child Academic Achievement: Math
Description: as for outcome 22
Time Frame: Age 8
Reporting Status: Not Posted, anticipated posting 2028-08

27. Primary Outcome: Child Fluid Reasoning
Description: Measured by the Wechsler Preschool and Primary Scale of Intelligence (WPPSI) fluid reasoning index, assessed through a composite of two tasks: picture concepts (score range: 0-27; higher scores indicate better performance) and matrix reasoning (score range: 0-26; higher scores indicate better performance). Expect higher scores in high- than low-cash gift group. Note: The Picture Concept subtest had to be dropped on 9/17/2024 due to floor effects.
  Reference:
  Wechsler, D. (2012). Wechsler Preschool and Primary Scale of Intelligence Fourth Edition (WPPSI-IV). San Antonio, TX: The Psychological Corporation.
Time Frame: Age 6
Reporting Status: Not Posted, anticipated posting 2026-08

28. Primary Outcome: Child Perceptual Reasoning
Description: Measured by the Wechsler Abbreviated Scale of Intelligence-Second Edition (WASI-II) perceptual reasoning index, assessed through a composite of two tasks: block design (score range: up to 8 years old: 0-57; > 9 yo: 0-71; higher scores indicate better performance) and matrix reasoning (up to 8 years old: 0-24; > 9 yo: 0-30; higher scores indicate better performance). Expect higher scores in high- than low-cash gift group.
  Reference:
  Wechsler, D. (2011). Wechsler Abbreviated Scale of Intelligence-Second Edition (WASI-II). San Antonio, TX: NCS Pearson.
Time Frame: Age 8
Reporting Status: Not Posted, anticipated posting 2028-08

29. Primary Outcome: Child Physiological Stress: Nail Cortisol
Description: Child nail samples will be collected to yield a measure of the concentration of cortisol in pg/mg (picograms per milligram). To ensure cortisol levels are within an expected range, values above 500 and equal to or less than 0 will be assigned a missing value. To account for potential outliers, values below 500 will be truncated at the 99th percentile. Cortisol values will be log-transformed. We hypothesize the high-cash gift group will have lower cortisol values when compared to the low-cash gift group. If both fingernail and toenail are collected we will control for whether fingernail or toenail.
  Reference: Phillips, R., Kraeuter, A. K., McDermott, B., Lupien, S., & Sarnyai, Z. (2021). Human nail cortisol as a retrospective biomarker of chronic stress: A systematic review. Psychoneuroendocrinology, 123, 104903.
Time Frame: Age 6
Reporting Status: Not Posted, anticipated posting 2026-08

30. Primary Outcome: Child Physiological Stress: Nail Cortisol
Description: as for outcome 29
Time Frame: Age 8
Reporting Status: Not Posted, anticipated posting 2028-08

31. Primary Outcome: Maternal Attentional Resources
Description: NIH Toolbox Flanker Inhibitory Control and Attention Test. Age-corrected standardized score. We expect a higher value of the maternal Flanker score for the high-cash gift group than the low-cash gift mothers. Higher scores indicate better performance. Prior to the Flanker administration, respondent/mother will be asked to listen and reflect for a minute on these questions: "Imagine that an unforeseen event requires of you an immediate $1,000 expense. Are there ways in which you may be able to come up with that amount of money on a very short notice? How would you go about it? How stressful would it be to manage this?
  Gershon et al. (2013). NIH Toolbox for assessment of neurological and behavioral function. Neurology, 80(11 Suppl 3) S2-S6.
  Slotkin J, et al. (2012) NIH Toolbox Scoring and Interpretation Guide (Northwestern and NIH).
  Zelazo PD, et al. (2013) II. NIH Toolbox cognition battery (CB): Measuring executive function and attention. Monogr Soc Res Child Dev 78:16-33.
Time Frame: Age 6
Reporting Status: Not Posted, anticipated posting 2026-08

32. Primary Outcome: Maternal Attentional Resources
Description: as for outcome 31
Time Frame: Age 8
Reporting Status: Not Posted, anticipated posting 2028-08

33. Secondary Outcome: Child Language Development: Language Milestones
Description: Language Milestones measured by Ages and Stages Questionnaire (ASQ)- Communication Subscale.
  We will estimate the statistical significance of the entire family of related measures in the Child Language Development outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Squires, J., Bricker, D. D., & Twombly, E. (2009). Ages & stages questionnaires. Baltimore, MD: Paul H. Brookes.
Time Frame: Age 12 months
Reporting Status: Not Posted

34. Secondary Outcome: Child Language Development: Vocabulary
Description: Communicative Development measured by Short Form Versions of MacArthur Communicative Development Inventories.
  We will estimate the statistical significance of the entire family of related measures in the Child Language Development outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Fenson, L. (2000). Short-form versions of the MacArthur Communicative Development Inventories. Applied Psycholinguistics, 21, 95 - 116.
Time Frame: Age 24 months
Reporting Status: Not Posted

35. Secondary Outcome: Child Executive Function: Executive Function
Description: Measured by the pencil tap test. This item was dropped on September 13, 2022, due to evidence of floor effects, and consistent reports from research staff that children were not understanding the instructions.
  Minimum value: 0; Maximum value: 16. Higher score indicates a better outcome.
  References:
  Diamond, A., & Taylor, C. (1996). Development of an aspect of executive control: development of the abilities to remember what I said and to "do as I say, not as I do". Developmental psychobiology, 29(4), 315-334.
Time Frame: Age 48 months
Reporting Status: Not Posted

36. Secondary Outcome: Child Socio-Emotional Processing: Behavior
Description: Behavior measured by NICHD Study of Early Child Care and Youth Development Mother-Child Interaction Task (positive/negative mood, activity level, sustained attention, positive engagement). Due to funding limitations, this was not feasible to code.
  Reference:
  Griffin, J. A., et al. (2007). NICHD Study of Early Childcare and Youth Development. National Institute of Health. Adapted script from mother-child-interaction at 15 months.
Time Frame: Age 12 months
Reporting Status: Not Posted

37. Secondary Outcome: Child Socio-Emotional Processing: Problems
Description: Problems measured by Brief Infant-Toddler Social and Emotional Assessment (BITSEA)- Problem Scale.
  Reference:
  Briggs-Gowan, M. J., Carter, A. S., Irwin, J. R., Wachtel, K., & Cicchetti, D. V. (2004). The Brief Infant-Toddler Social and Emotional Assessment: screening for social-emotional problems and delays in competence. Journal of pediatric psychology, 29(2), 143-155.
Time Frame: Age 12 months
Reporting Status: Not Posted

38. Secondary Outcome: Child Socio-Emotional Processing: Problems
Description: Problems measured by Brief Infant-Toddler Social and Emotional Assessment (BITSEA).
  We will estimate the statistical significance of the family of related measures in the Child Socio-Emotional Processing outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Briggs-Gowan, et al. (2004). The Brief Infant-Toddler Social and Emotional Assessment: screening for social-emotional problems and delays in competence. Journal of pediatric psychology, 29(2), 143-155.
Time Frame: Age 24 months
Reporting Status: Not Posted

39. Secondary Outcome: Child Pre-Literacy
Description: Pre-Literacy measured by The Reading House.
  Minimum value: 0; Maximum value: 14. Higher score indicates a better outcome.
  Reference:
  Hutton, et al. (2019). The Reading House: A Children's Book for Emergent Literacy Screening During Well-Child Visits. Pediatrics, 143 (6): e20183843. 10.1542/peds.2018-3843
  Hutton et al. (2021). Validation of The Reading House and Association With Cortical Thickness. Pediatrics, 147(3), e20201641. https://doi.org/10.1542/peds.2020-1641
Time Frame: Age 48 months
Reporting Status: Not Posted

40. Secondary Outcome: Child Intelligence Quotient
Description: Measured by the Wechsler Nonverbal Scale of Ability. Modified on September 30, 2022 to no longer measure child IQ, as described below.
  Minimum score: 10; Maximum score: 90. Higher score indicates a better outcome.
  Note: The IQ score is calculated using two subtests -- Matrices and Recognition -- and we began our fieldwork on July 9, 2022 with both. On the basis of preliminary analysis of the first 71 cases, we discovered that 21% of participants scored at the floor of the Recognition assessment. We therefore dropped the Recognition subtest from our data collection instrument on September 30 2022, precluding us from calculating IQ in subsequent participants. Scores on the Matrices subtest, which measures visual processing and abstract spatial perception (not IQ per se), are now registered as an age-4 secondary outcome.
  Reference:
  Wechsler, D., Naglieri, J. A. (2006). Wechsler Nonverbal Scale of Ability. San Antonio, TX: Pearson.
Time Frame: Age 48 months
Reporting Status: Not Posted

41. Secondary Outcome: Child Resting Brain Function
Description: Measured by EEG
  We will estimate the statistical significance of the entire family of related measures in the Child Brain Function outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  References:
  Tomalski, P., Moore, D. G., Ribeiro, H., Axelsson, E. L., Murphy, E., Karmiloff-Smith, A., ... & Kushnerenko, E. (2013). Socioeconomic status and functional brain development-associations in early infancy. Developmental Science, 16(5), 676-687.
  Otero, G. A., Pliego-Rivero, F. B., Fernández, T., & Ricardo, J. E. E. G. (2003). EEG development in children with sociocultural disadvantages: a follow-up study. Clinical neurophysiology, 114(10), 1918-1925.
  Marshall, P. J., Fox, N. A., & Group, B. C. (2004). A comparison of the electroencephalogram between institutionalized and community children in Romania. Journal of Cognitive Neuroscience, 16(8), 1327-1338.
Time Frame: Age 12 months
Reporting Status: Not Posted

42. Secondary Outcome: Child Resting Brain Function
Description: Measured by EEG.
  We hypothesize greater frontal gamma power in the high-cash gift group, and plan to analyze a full model of regions nested within bands, with the plan to report all exploratory outcomes. See analysis plan.
  References:
  Tomalski, P., et al. (2013); Otero, G. A., et. al (2003); Marshall, P. J., et.al. (2004)
  Troller-Renfree, S. V., et. al. (2022). The impact of a poverty reduction intervention on infant brain activity. Proceedings of the National Academy of Sciences, 119(5).
Time Frame: Age 48 months
Reporting Status: Not Posted

43. Secondary Outcome: Child Resting Brain Function
Description: Our primary hypothesis (detailed above) is based on data gathered in the eyes- closed condition. We also preregister the corresponding analyses of data from the eyes-open condition as secondary hypotheses, with the same directional hypotheses as the eyes-closed condition. A second set of secondary analyses are based on a different estimation approach. Consistent with another RCT examining brain activity, we will analyze band-specific effects using mixed-effects models, with group as the between-subjects factor and region as within-subjects factor, to examine ITT impacts on each band of relative power in the eyes-closed condition. Our secondary hypotheses for each band are as follows: Theta (high-cash<low-cash), Alpha (high-cash>low-cash), Beta (high-cash>low-cash), and Gamma (high-cash>low-cash). One-tailed t-tests will be used given directional hypotheses. No further multiple-testing adjustments beyond the us use of multi-level models will be used. See Statistical Analysis Plan.
Time Frame: Age 6
Reporting Status: Not Posted

44. Secondary Outcome: Child Resting Brain Function
Description: as for outcome 43
Time Frame: Age 8
Reporting Status: Not Posted

45. Secondary Outcome: Child Task-Related Brain Function
Description: Auditory Discrimination Brain Function measured by mismatch negativity (MMN) ERP with larger differences between standard and deviant stimulus in high-cash gift group compared to the low-cash gift group.
  References:
  Cheour, M., Leppänen, P. H., & Kraus, N. (2000). Mismatch negativity (MMN) as a tool for investigating auditory discrimination and sensory memory in infants and children. Clinical neurophysiology, 111(1), 4-16.
  Garcia-Sierra, A., et al.. (2011). Bilingual language learning: An ERP study relating early brain responses to speech, language input, and later word production. Journal of Phonetics, 39(4), 546-557.
  Kuhl, P. K., et al.. (2005). Links between social and linguistic processing of speech in preschool children with autism: behavioral and electrophysiological measures. Developmental science, 8(1), F1-F12.
Time Frame: Age 48 months
Reporting Status: Not Posted

46. Secondary Outcome: Child Health: Body Mass Index (BMI)
Description: Measured by CDC BMI percentage scales.
  Reference:
  Kuczmarski, R. J. (2000). CDC growth charts; United States.
Time Frame: Age 48 months
Reporting Status: Not Posted

47. Secondary Outcome: Child Health: Body Mass Index (BMI)
Description: Body Mass Index. Measured by CDC BMI percentile scales. We expect to see a reduced percentage of overweight or obese (greater than or equal to 85th percentile) children in the high-cash gift group compared to the low-cash gift group. We will report mean percentile scores of the two groups in descriptive analyses.
Time Frame: Age 6
Reporting Status: Not Posted

48. Secondary Outcome: Child Health: Body Mass Index (BMI)
Description: as for outcome 47
Time Frame: Age 8
Reporting Status: Not Posted

49. Secondary Outcome: Child Health, Physiological Stress
Description: Measured by hair cortisol concentration.
  Note: Our original plan was to measure physiological stress using hair cortisol concentration. The first several months of data collection revealed large racial and ethnic differences in willingness to provide a hair sample, due to both cultural and practical reasons. Because of the large amounts of non-random missing data, which would both compromise our statistical power and limit the generalizability of any findings, we dropped hair cortisol from our data collection procedures on October 25, 2022.
  Reference:
  Ursache, A., Merz, E. C., Melvin, S., Meyer, J., & Noble, K. G. (2017). Socioeconomic status, hair cortisol and internalizing symptoms in parents and children. Psychoneuroendocrinology, 78, 142-150.
Time Frame: Age 48 months
Reporting Status: Not Posted

50. Secondary Outcome: Child Health, Sleep
Description: Measured by an adapted Short Form of Patient-Reported Outcomes Measurement Information System (PROMIS™)
  Minimum score: 4; Maximum score: 20. Higher score indicates a better outcome.
  Reference:
  Yu, L., Buysse, D. J., Germain, A., Moul, D. E., Stover, A., Dodds, N. E., ... & Pilkonis, P. A. (2012). Development of short forms from the PROMIS™ sleep disturbance and sleep-related impairment item banks. Behavioral sleep medicine, 10(1), 6-24.
Time Frame: Age 12 Months
Reporting Status: Not Posted

51. Secondary Outcome: Child Health, Sleep
Description: as for outcome 50
Time Frame: Age 24 months
Reporting Status: Not Posted

52. Secondary Outcome: Child Health, Overall Health, Medical Care, Diagnosis of Condition or Disability
Description: Measured by an index of six items (see Appendix Table 7 in "Analysis Plan and Measures" document for items)
  Reference:
  Halim, M. L., Yoshikawa, H., & Amodio, D. M. (2013). Cross-generational effects of discrimination among immigrant mothers: Perceived discrimination predicts child's healthcare visits for illness. Health Psychology, 32(2), 203.
Time Frame: Age 12 months
Reporting Status: Not Posted

53. Secondary Outcome: Child Health, Overall Health, Medical Care, Diagnosis of Condition or Disability
Description: as for outcome 52
Time Frame: Age 24 months
Reporting Status: Not Posted

54. Secondary Outcome: Child Health, Overall Health, Diagnosis of Condition or Disability
Description: Measured by an index of survey items (see Appendix Table 7 in "Analysis Plan and Measures" document for items).
  Reference:
  Idler, E. L., & Benyamini, Y. (1997). Self-rated health and mortality: a review of twenty-seven community studies. Journal of health and social behavior, 21-37
Time Frame: Age 48 months
Reporting Status: Not Posted

55. Secondary Outcome: Child Health, Overall Health
Description: Measured by an index of survey items (see Appendix Table 9 in "Analysis Plan and Measures" document for items).
  Reference:
  Idler, E. L., & Benyamini, Y. (1997). Self-rated health and mortality: a review of twenty-seven community studies. Journal of health and social behavior, 21-37
Time Frame: Age 6
Reporting Status: Not Posted

56. Secondary Outcome: Child Health, Overall Health
Description: as for outcome 55
Time Frame: Age 8
Reporting Status: Not Posted

57. Secondary Outcome: Child Health: Chronic Health Condition
Description: Has child been diagnosed with any chronic health condition? Yes/No. If yes; asthma and/or something else. Expect lower rate in high- than low-cash gift group.
  Reference: BFY Study PIs
Time Frame: Age 6
Reporting Status: Not Posted

58. Secondary Outcome: Child Health: Chronic Health Condition
Description: as for outcome 57
Time Frame: Age 8
Reporting Status: Not Posted

59. Secondary Outcome: Child Epigenetic Pace of Aging
Description: Measured using method reported in Appendix Table 7 in "Analysis Plan and Measures" document. Please also see preregistration at OSF: https://osf.io/ahv2p/?view_only=
  Reference:
  Belsky, W. D. et al. (2020). Quantification of the pace of biological aging in humans through blood test, the DunedinPoAm DNA methylation algorithm. eLife 9:e54870. https://doi.org/10.7554/eLife.54870
  Belsky, W. D. et al. (2022). DunedinPACE, a DNA methylation biomarker of the pace of aging. eLife 11:e73420. https://doi.org/10.7554/eLife.73420
Time Frame: Age 48 months
Reporting Status: Not Posted

60. Secondary Outcome: Child Epigenetic Pace of Aging
Description: Methylation pace of aging was developed from DNA-methylation analysis of Pace of Aging in the Dunedin Study birth cohort. Pace of Aging is a composite phenotype derived from analysis of longitudinal change in 18 biomarkers of organ-system integrity. In contrast, so-called epigenetic clocks are trained on chronological age. Increments of methylation pace of aging correspond to "years" of physiological change occurring per 12-months of chronological time. The second iteration (DunedinPACE) takes into account an additional measurement occasion and only includes the most reliable DNA methylation probes, i.e. probes with little variation between technical replicates. If a higher quality measure of epigenetic aging at the time of analysis becomes available, we we will substitute that instead.We will also report GrimAge Acceleration, which we consider an exploratory analysis. GrimAge represents a DNA-methylation metric designed to predict morbidity and mortality.
  References: see Table 9
Time Frame: Age 6
Reporting Status: Not Posted

61. Secondary Outcome: Child Epigenetic Pace of Aging
Description: as for outcome 60
Time Frame: Age 8
Reporting Status: Not Posted

62. Secondary Outcome: Child DNA Methylation
Description: Measured using method reported in Appendix Table 7 in "Analysis Plan and Measures" document. Please also see preregistration at OSF: https://osf.io/ahv2p/?view_only=
  Reference:
  McCartney, D.L., Hillary, R.F., Conole, E.L.S. et al. Blood-based epigenome-wide analyses of cognitive abilities. Genome Biol 23, 26 (2022). https://doi.org/10.1186/s13059-021-02596-5
Time Frame: Age 48 months
Reporting Status: Not Posted

63. Secondary Outcome: Child DNA Methylation
Description: Salivary DNA-methylation profiles of cognitive functioning, i.e., "Epigenetic-g", can be computed on the basis of weights from a blood-based epigenome wide association study of general cognitive functions (g) in adults (McCartney et al., 2022). General cognitive ability was derived from the first unrotated principal component of logical memory, verbal fluency and digit symbol tests, and vocabulary. Epigenetic-g is conceptually distinct from biological aging. If a higher quality measure of epigenetic profile of cognitive functioning becomes available at the time of analysis, we we will substitute that instead.
  Reference: McCartney, D.L., Hillary, R.F., Conole, E.L.S. et al. Blood-based epigenome-wide analyses of cognitive abilities. Genome Biol 23, 26 (2022). https://doi.org/10.1186/s13059-021-02596-5
Time Frame: Age 6
Reporting Status: Not Posted

64. Secondary Outcome: Child DNA Methylation
Description: as for outcome 63
Time Frame: Age 8
Reporting Status: Not Posted

65. Secondary Outcome: Child Nutrition: Consumption of Healthy Foods
Description: Measured by an index of survey items (see Appendix Table 7 in "Analysis Plan and Measures" document for items).
  Reference:
  Los Angeles County WIC Survey. (2017). Retrievable from: http://lawicdata.org/wp-content/uploads/2014/09/WIC-Parents-Quex-English-FINAL.pdf
Time Frame: Age 24 months
Reporting Status: Not Posted

66. Secondary Outcome: Child Nutrition: Consumption of Healthy Food
Description: Measured by an index of survey items (see Appendix Table 9 in "Analysis Plan and Measures" document for items).
  Expect higher scores in high- than low-cash gift group.
  Reference:
  Los Angeles County WIC Survey. (2017). Retrievable from: http://lawicdata.org/wp-content/uploads/2014/09/WIC-Parents-Quex-English-FINAL.pdf
Time Frame: Age 6
Reporting Status: Not Posted

67. Secondary Outcome: Child Nutrition: Consumption of Healthy Foods
Description: as for outcome 66
Time Frame: Age 8
Reporting Status: Not Posted

68. Secondary Outcome: Child Nutrition: Consumption of Unhealthy Foods
Description: as for outcome 65
Time Frame: Age 24 months
Reporting Status: Not Posted

69. Secondary Outcome: Child Nutrition: Consumption of Unhealthy Foods
Description: Measured by an index of survey items (see Appendix Table 9 in "Analysis Plan and Measures" document for items).
  Expect lower scores in high- than low-cash gift group.
  References:
  Los Angeles County WIC Survey. (2017). Retrievable from: http://lawicdata.org/wp-content/uploads/2014/09/WIC-Parents-Quex-English-FINAL.pdf Hunsberger M, O'Malley J, Block T, Norris JC. Relative validation of Block Kids Food Screener for dietary assessment in children and adolescents. Matern Child Nutr. 2012:1-11. doi:10.1111/j.1740-8709.2012.00446.x.
Time Frame: Age 6
Reporting Status: Not Posted

70. Secondary Outcome: Child Nutrition: Consumption of Unhealthy Foods
Description: as for outcome 69
Time Frame: Age 8
Reporting Status: Not Posted

71. Secondary Outcome: Any Maternal Concern for Developmental Delay: Total "Predictive Concerns" in the Parents' Evaluation of Developmental Status (PEDS)
Description: Measured by the total number of maternal-reported concerns that are "predictive of developmental delay" in the Parents' Evaluation of Developmental Status (PEDS).
  Minimum score: 0; Maximum score: 5. Higher score indicates worse outcome.
  We will estimate the statistical significance of the entire family of related measures in the Any Maternal Concern for Developmental Delay outcome cluster using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Glascoe FP. Parents' Evaluations of Developmental Status: A Method for Detecting and Addressing Developmental and Behavioral Problems in Children. Nashville, TN: Ellsworth & Vandermeer Press, 1997.
Time Frame: Age 36 months
Reporting Status: Not Posted

72. Secondary Outcome: Any Maternal Concern for Developmental Delay: Parents' Evaluation of Developmental Status (PEDS)
Description: Measured by the total score across categories of components of the Parents' Evaluation of Developmental Status (PEDS), which includes 10 survey items.
  Minimum score: 0; Maximum score: 10. Higher score indicates worse outcome.
  We will estimate the statistical significance of the entire family of related measures in the Any Maternal Concern for Developmental Delay outcome cluster using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Glascoe FP. Parents' Evaluations of Developmental Status: A Method for Detecting and Addressing Developmental and Behavioral Problems in Children. Nashville, TN: Ellsworth & Vandermeer Press, 1997.
Time Frame: Age 36 months
Reporting Status: Not Posted

73. Secondary Outcome: Diagnosis of Developmental Condition
Description: Measured by one dichotomous survey item (see Appendix Table 7 in "Analysis Plan and Measures" document for items).
  Minimum score: 0; Maximum score: 1. Higher score indicates a worse outcome.
  Reference:
  Study PIs
Time Frame: Age 48 months
Reporting Status: Not Posted

74. Secondary Outcome: Diagnosis of Developmental Condition
Description: Dichotomous measure 1:yes 0:no, constructed from the questionnaire categories: Diagnosis of Dev. Condition: speech delay, autism, ADHD, something else (this Q is part of Health Qs) We will estimate whether there are group differences, but do not formulate a directional hypothesis, because of two offsetting possibilities: i) the high-cash gift group may have better access to services, which may lead to higher rates of diagnosis and/or ii) the cash gifts may lead to fewer developmental conditions
Time Frame: Age 6
Reporting Status: Not Posted

75. Secondary Outcome: Diagnosis of Developmental Condition
Description: as for outcome 74
Time Frame: Age 8
Reporting Status: Not Posted

76. Secondary Outcome: Child Special Services (IEP)
Description: Maternal report of whether the child has an IEP or receives special educational services using questions adapted from the School Enrollment and Expectations section of the PSID Child Development Supplement. 1: yes; 0: no We will estimate whether there are group differences, but do not formulate a directional hypothesis, because of two offsetting possibilities: i) the high-cash gift group may have better access to services, which may lead to higher rates of diagnosis and receipt of special education and/or ii) the cash gifts may lead to higher school achievement and therefore lower need for special education and individual education plans.
  Reference: Adapted from the School Enrollment and Expectations (SEE) section of the 2021 Panel Study of Income Dynamics (PSID) Child Development Supplement: Beaule et al.(2023). PSID-2021 Main Interview User Manual: Release 2023. Institute
Time Frame: Age 6
Reporting Status: Not Posted

77. Secondary Outcome: Child Special Services (IEP)
Description: as for outcome 76
Time Frame: Age 8
Reporting Status: Not Posted

78. Secondary Outcome: Household Economic Hardship: Household Poverty Rate
Description: Household Poverty Rate measured using the Census Bureau's Poverty thresholds by Size of Family and Number of Children.
  We will estimate the statistical significance of the entire family of related measures in the Household Economic Hardship outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  US Census Bureau
Time Frame: Age 12 months
Reporting Status: Not Posted

79. Secondary Outcome: Household Economic Hardship: Household Poverty Rate
Description: as for outcome 78
Time Frame: Age 24 months
Reporting Status: Not Posted

80. Secondary Outcome: Household Economic Hardship: Household Poverty Rate
Description: as for outcome 78
Time Frame: Age 36 months
Reporting Status: Not Posted

81. Secondary Outcome: Household Economic Hardship: Household Poverty Rate
Description: as for outcome 78
Time Frame: Age 48 months
Reporting Status: Not Posted

82. Secondary Outcome: Household Economic Hardship: Household Poverty Rate
Description: as for outcome 78
Time Frame: Age 6
Reporting Status: Not Posted

83. Secondary Outcome: Household Economic Hardship: Household Poverty Rate
Description: as for outcome 78
Time Frame: Age 8
Reporting Status: Not Posted

84. Secondary Outcome: Household Economic Hardship: Index of Economic Stress
Description: Index of Economic Stress measured by an additive index of nine items (see Appendix Table 8 in "Analysis Plan and Measures" document for items).
  We will estimate the statistical significance of the entire family of related measures in the Household Economic Hardship outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Kling, J.R., Liebman, J.B., Katz, L.F. (2007). Experimental analysis of neighborhood effects. Econometrica, 75(1), 83-119.
Time Frame: Age 12 months
Reporting Status: Not Posted

85. Secondary Outcome: Household Economic Hardship: Index of Economic Stress
Description: as for outcome 84
Time Frame: Age 24 months
Reporting Status: Not Posted

86. Secondary Outcome: Household Economic Hardship: Index of Economic Stress
Description: Index of Economic Stress measured by an additive index of nine items (see Appendix Table 8 in "Analysis Plan and Measures" document for items).
  Minimum score: 0; Maximum score: 9. Higher score indicates worse outcome.
  We will estimate the statistical significance of the entire family of related measures in the Household Economic Hardship outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Kling, J.R., Liebman, J.B., Katz, L.F. (2007). Experimental analysis of neighborhood effects. Econometrica, 75(1), 83-119.
Time Frame: Age 36 months
Reporting Status: Not Posted

87. Secondary Outcome: Household Economic Hardship: Index of Economic Stress
Description: as for outcome 86
Time Frame: Age 48 months
Reporting Status: Not Posted

88. Secondary Outcome: Household Economic Hardship: Index of Ecomomic Stress
Description: Index of Economic Stress measured by an additive index of six items (see Appendix Table 10 in "Analysis Plan and Measures" document for items).
  Minimum score: 0; Maximum score: 6. Higher score indicates more ecomomic stress. Expect less stress for high-cash group.
  We will estimate the statistical significance of the entire family of related measures in the Household Economic Hardship outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Kling, J.R., Liebman, J.B., Katz, L.F. (2007). Experimental analysis of neighborhood effects. Econometrica, 75(1), 83-119.
Time Frame: Age 6
Reporting Status: Not Posted

89. Secondary Outcome: Household Economic Hardship: Index of Economic Stress
Description: as for outcome 88
Time Frame: Age 8
Reporting Status: Not Posted

90. Secondary Outcome: Household Economic Hardship: Maternal Hardship
Description: Maternal Hardship measured by one item (see Appendix Table 10 in "Analysis Plan and Measures" document).
  Minimum score: 1; Maximum score: 4. Higher score indicates more hardship. Expect less hardship for high-cash group.
  We will estimate the statistical significance of the entire family of related measures in the Household Economic Hardship outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference: BFY Study PIs
Time Frame: Age 6
Reporting Status: Not Posted

91. Secondary Outcome: Household Economic Hardship: Maternal Hardship
Description: as for outcome 90
Time Frame: Age 8
Reporting Status: Not Posted

92. Secondary Outcome: Household Economic Hardship: Index of Food Insecurity
Description: Index of Food Insecurity measured by the U.S. Household Food Security Survey Module: Six-Item Short Form.
  We will estimate the statistical significance of the entire family of related measures in the Household Economic Hardship outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  The U.S. Household Food Security Survey Module: Six-Item Short Form retrieved from: https://www.ers.usda.gov/media/8282/short2012.pdf
Time Frame: Age 12 months
Reporting Status: Not Posted

93. Secondary Outcome: Household Economic Hardship: Index of Food Insecurity
Description: as for outcome 92
Time Frame: Age 24 months
Reporting Status: Not Posted

94. Secondary Outcome: Household Economic Hardship: Index of Food Insecurity
Description: as for outcome 92
Time Frame: Age 36 months
Reporting Status: Not Posted

95. Secondary Outcome: Household Economic Hardship: Index of Food Insecurity
Description: as for outcome 92
Time Frame: Age 48 months
Reporting Status: Not Posted

96. Secondary Outcome: Social Services Receipt; Number of Benefits Received by Mother
Description: Measured by an additive index of 9 items (see Appendix Table 8 in "Analysis Plan and Measures" document for items).
  Reference: study PIs
Time Frame: Age 12 months
Reporting Status: Not Posted

97. Secondary Outcome: Social Services Receipt; Number of Benefits Received by Mother
Description: as for outcome 96
Time Frame: Age 24 months
Reporting Status: Not Posted

98. Secondary Outcome: Social Services Receipt; Number of Benefits Received by Mother
Description: Measured by an additive index of 9 items (see Appendix Table 8 in "Analysis Plan and Measures" document for items).
  Minimum score: 0; Maximum score: 5.
  Reference: study PIs
Time Frame: Age 36 months
Reporting Status: Not Posted

99. Secondary Outcome: Mother's Labor Market and Education Participation: Time to Labor Market Re-entry From Birth
Description: Time to Labor Market Re-entry from Birth measured by the number of months from child's birth until mother's reentry into the labor market (see Appendix Table 8 in "Analysis Plan and Measures" document for items).
  We will estimate the statistical significance of the entire family of related measures in the Mother's Labor Market and Education Participation outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference: study PIs
Time Frame: Age 12 months
Reporting Status: Not Posted

100. Secondary Outcome: Mother's Labor Market and Education Participation: Time to Full-Time Labor Market Reentry From Birth
Description: Time to Full-Time Labor Market Reentry from Birth measured by the number of months from child's birth until mother's full-time reentry into the labor market (see Appendix Table 8 in "Analysis Plan and Measures" document for items).
  We will estimate the statistical significance of the entire family of related measures in the Mother's Labor Market and Education Participation outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference: study PIs
Time Frame: Age 12 months
Reporting Status: Not Posted

101. Secondary Outcome: Mother's Labor Market and Education Participation: Mother's Labor Market Participation
Description: Dichotomous variable indicating whether mother is participating in the labor market.
  We will estimate the statistical significance of the entire family of related measures in the Mother's Labor Market and Education Participation outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference: BFY Study PIs
Time Frame: Age 48 months
Reporting Status: Not Posted

102. Secondary Outcome: Mother's Labor Market and Education Participation: Mother's Labor Market Participation
Description: as for outcome 101
Time Frame: Age 6
Reporting Status: Not Posted

103. Secondary Outcome: Mother's Labor Market and Education Participation: Mother's Labor Market Participation
Description: as for outcome 101
Time Frame: Age 8
Reporting Status: Not Posted

104. Secondary Outcome: Mother's Labor Market and Education Participation: Mother's Education and Training Attainment
Description: Mother's Education and Training Attainment measured by a survey item (see Appendix Table 8 in "Analysis Plan and Measures" document for items).
  We will estimate the statistical significance of the entire family of related measures in the Mother's Labor Market and Education Participation outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference: study PIs
Time Frame: Age 12 months
Reporting Status: Not Posted

105. Secondary Outcome: Mother's Labor Market and Education Participation: Mother's Education and Training Attainment
Description: as for outcome 104
Time Frame: Age 24 months
Reporting Status: Not Posted

106. Secondary Outcome: Mother's Labor Market and Education Participation: Mother's Education and Training Attainment
Description: Mother's Education and Training Attainment measured by a survey item (see Appendix Table 8 in "Analysis Plan and Measures" document for items).
  Minimum score: 0; Maximum score: 1. Higher score indicates better outcome.
  We will estimate the statistical significance of the entire family of related measures in the Mother's Labor Market and Education Participation outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference: study PIs
Time Frame: Age 36 months
Reporting Status: Not Posted

107. Secondary Outcome: Mother's Labor Market and Education Participation: Mother's Education Attainment
Description: Mother's Education Attainment measured by a survey item (see Appendix Table 10 in "Analysis Plan and Measures" document for items).
  Minimum score: 0; Maximum score: 1. Higher score indicates better outcome. Expect more education in high-cash gift group.
  We will estimate the statistical significance of the entire family of related measures in the Mother's Labor Market and Education Participation outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference: BFY Study PIs
Time Frame: Age 6
Reporting Status: Not Posted

108. Secondary Outcome: Mother's Labor Market and Education Participation: Mother's Education Attainment
Description: as for outcome 107
Time Frame: Age 8
Reporting Status: Not Posted

109. Secondary Outcome: Mother's Labor Market and Education Participation: Mother's Training Attainment
Description: Mother's Training Attainment measured by a survey item (see Appendix Table 10 in "Analysis Plan and Measures" document for items).
  Minimum score: 0; Maximum score: 1. Higher score indicates better outcome. Expect more training in high-cash gift group.
  We will estimate the statistical significance of the entire family of related measures in the Mother's Labor Market and Education Participation outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference: BFY Study PIs
Time Frame: Age 6
Reporting Status: Not Posted

110. Secondary Outcome: Mother's Labor Market and Education Participation: Mother's Training Attainment
Description: as for outcome 109
Time Frame: Age 8
Reporting Status: Not Posted

111. Secondary Outcome: Mother's Labor Market and Education Participation: Maternal Earnings
Description: Mother's Earnings in the previous calendar year
  We will estimate the statistical significance of the entire family of related measures in the Mother's Labor Market and Education Participation outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference: Panel Study of Income Dynamics (PSID)
Time Frame: Age 48 months
Reporting Status: Not Posted

112. Secondary Outcome: Mother's Labor Market and Education Participation: Maternal Earnings
Description: Mother's Earnings in the previous calendar year. Expect higher income for high-cash group.
  We will estimate the statistical significance of the entire family of related measures in the Mother's Labor Market and Education Participation outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference: Panel Study of Income Dynamics (PSID)
Time Frame: Age 6
Reporting Status: Not Posted

113. Secondary Outcome: Mother's Labor Market and Education Participation: Maternal Earnings
Description: as for outcome 112
Time Frame: Age 8
Reporting Status: Not Posted

114. Secondary Outcome: Child-Focused Expenditures: Index of Expenditures Since Birth
Description: Index of Child-Focused Expenditures since birth measured by an additive index of survey items (see Appendix Table 8 in "Analysis Plan and Measures" document for items).
  We will estimate the statistical significance of the entire family of related measures in the Child-Focused Expenditures outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Lugo-Gil, J., Yoshikawa, H. (2006). Assessing expenditures on children in low-income, ethnically diverse, and immigrant families. National Poverty Center Working Paper Series, 06-36.
  National Study of Early Care and Education
Time Frame: Age 12 months
Reporting Status: Not Posted

115. Secondary Outcome: Child-Focused Expenditures: Index of Expenditures in Past 30 Days
Description: Index of Expenditures in past 30 days measured by a dollar amount sum of responses to survey items (see Appendix Table 8 in "Analysis Plan and Measures" document for items).
  We will estimate the statistical significance of the entire family of related measures in the Child-Focused Expenditures outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Lugo-Gil, J., Yoshikawa, H. (2006). Assessing expenditures on children in low-income, ethnically diverse, and immigrant families. National Poverty Center Working Paper Series, 06-36.
  National Study of Early Care and Education
Time Frame: Age 12 months
Reporting Status: Not Posted

116. Secondary Outcome: Child-Focused Expenditures: Index of Expenditures in Past 30 Days
Description: Index of Expenditures in past 30 days measured by a dollar amount sum of responses to survey items (see Appendix Table 8 in "Analysis Plan and Measures" document for items).
  We will estimate the statistical significance of the entire family of related measures in the Child-Focused Expenditures outcome cluster using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Lugo-Gil, J., Yoshikawa, H. (2006). Assessing expenditures on children in low-income, ethnically diverse, and immigrant families. National Poverty Center Working Paper Series, 06-36.
  National Study of Early Care and Education
Time Frame: Age 24 months
Reporting Status: Not Posted

117. Secondary Outcome: Child-Focused Expenditures: Index of Expenditures in Past 30 Days
Description: Index of Expenditures in past 30 days measured by a dollar amount sum of responses to survey items (see Appendix Table 8 in "Analysis Plan and Measures" document for items).
  Higher score indicates better outcome.
  We will estimate the statistical significance of the entire family of related measures in the Child-Focused Expenditures outcome cluster using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Lugo-Gil, J., Yoshikawa, H. (2006). Assessing expenditures on children in low-income, ethnically diverse, and immigrant families. National Poverty Center Working Paper Series, 06-36.
  National Study of Early Care and Education
Time Frame: Age 36 months
Reporting Status: Not Posted

118. Secondary Outcome: Child-Focused Expenditures: Index of Expenditures in Past 30 Days
Description: as for outcome 115
Time Frame: Age 48 months
Reporting Status: Not Posted

119. Secondary Outcome: Child-focused Expenditures: Index of Child-Focused Expenditures in Past 30 Days
Description: Index of Expenditures in past 30 days measured by a dollar amount sum of responses to survey items (see Appendix Table 10 in "Analysis Plan and Measures" document for items). Expect higher spending for high-cash group.
  We will estimate the statistical significance of the entire family of related measures in the Child-Focused Expenditures outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  References:
  Lugo-Gil, J., Yoshikawa, H. (2006). Assessing expenditures on children in low-income, ethnically diverse, and immigrant families. National Poverty Center Working Paper Series, 06-36.
  Schild et al. (2023). Effects of the Expanded Child Tax Credit on Household Spending: Estimates Based on US Consumer Expenditure Survey Data (No. w31412). National Bureau of Economic Research. https://www.bls.gov/osmr/research-papers/2023/pdf/ec230010.pdf
Time Frame: Age 6
Reporting Status: Not Posted

120. Secondary Outcome: Child-focused Expenditures: Index of Child-focused Expenditures in Past 30 Days
Description: as for outcome 119
Time Frame: Age 8
Reporting Status: Not Posted

121. Secondary Outcome: Child-focused Expenditures: Index of Expenditures on All Children in the Household, Including Target Child
Description: as for outcome 119
Time Frame: Age 6
Reporting Status: Not Posted

122. Secondary Outcome: Child-focused Expenditures: Index of Expenditures on All Children in the Household, Including Target Child
Description: as for outcome 119
Time Frame: Age 8
Reporting Status: Not Posted

123. Secondary Outcome: Child-Focused Expenditures: Cost of Paid Child Care
Description: Cost of Paid Child Care measured by survey item (see Appendix Table 8 in "Analysis Plan and Measures" document for items).
  We will estimate the statistical significance of the entire family of related measures in the Child-Focused Expenditures outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Lugo-Gil, J., Yoshikawa, H. (2006). Assessing expenditures on children in low-income, ethnically diverse, and immigrant families. National Poverty Center Working Paper Series, 06-36.
  National Study of Early Care and Education
Time Frame: Age 12 months
Reporting Status: Not Posted

124. Secondary Outcome: Child-Focused Expenditures: Cost of Paid Child Care
Description: Cost of Paid Child Care measured by survey item (see Appendix Table 8 in "Analysis Plan and Measures" document for items).
  We will estimate the statistical significance of the entire family of related measures in the Child-Focused Expenditures outcome cluster using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Lugo-Gil, J., Yoshikawa, H. (2006). Assessing expenditures on children in low-income, ethnically diverse, and immigrant families. National Poverty Center Working Paper Series, 06-36.
  National Study of Early Care and Education
Time Frame: Age 24 months
Reporting Status: Not Posted

125. Secondary Outcome: Child-Focused Expenditures: Cost of Paid Child Care
Description: Cost of Paid Child Care measured by survey item (see Appendix Table 8 in "Analysis Plan and Measures" document for items).
  Higher score indicates better outcome.
  We will estimate the statistical significance of the entire family of related measures in the Child-Focused Expenditures outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Lugo-Gil, J., Yoshikawa, H. (2006). Assessing expenditures on children in low-income, ethnically diverse, and immigrant families. National Poverty Center Working Paper Series, 06-36.
  National Study of Early Care and Education
Time Frame: Age 36 months
Reporting Status: Not Posted

126. Secondary Outcome: Child-Focused Expenditures: Cost of Paid Child Care
Description: as for outcome 125
Time Frame: Age 48 months
Reporting Status: Not Posted

127. Secondary Outcome: Child-Focused Expenditures: Use of Center-Based Care
Description: Use of Center-Based Care measured by survey item (see Appendix Table 8 in "Analysis Plan and Measures" document for items).
  We will estimate the statistical significance of the entire family of related measures in the Child-Focused Expenditures outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Lugo-Gil, J., Yoshikawa, H. (2006). Assessing expenditures on children in low-income, ethnically diverse, and immigrant families. National Poverty Center Working Paper Series, 06-36.
  National Study of Early Care and Education
Time Frame: Age 12 months
Reporting Status: Not Posted

128. Secondary Outcome: Child-Focused Expenditures: Use of Center-Based Care
Description: as for outcome 127
Time Frame: Age 24 months
Reporting Status: Not Posted

129. Secondary Outcome: Child-Focused Expenditures: Use of Center-Based Care
Description: Use of Center-Based Care measured by survey item (see Appendix Table 8 in "Analysis Plan and Measures" document for items).
  Minimum score: 0; Maximum score: 1. Higher score indicates better outcome.
  We will estimate the statistical significance of the entire family of related measures in the Child-Focused Expenditures outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Lugo-Gil, J., Yoshikawa, H. (2006). Assessing expenditures on children in low-income, ethnically diverse, and immigrant families. National Poverty Center Working Paper Series, 06-36.
  National Study of Early Care and Education
Time Frame: Age 48 months
Reporting Status: Not Posted

130. Secondary Outcome: Child-Focused Expenditures: Use of Center-Based Care
Description: as for outcome 129
Time Frame: Age 36 months
Reporting Status: Not Posted

131. Secondary Outcome: Housing and Neighborhoods: Index of Perceptions of Neighborhood Safety
Description: Index of Perceptions of Neighborhood Safety measured by an additive index of survey items (see Appendix Table 8 in "Analysis Plan and Measures" document for items).
  We will estimate the statistical significance of the entire family of related measures in the Housing and Neighborhoods outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Kling, J.R., Liebman, J.B., Katz, L.F. (2007). Experimental analysis of neighborhood effects. Econometrica, 75(1), 83-119.
Time Frame: Age 12 months
Reporting Status: Not Posted

132. Secondary Outcome: Housing and Neighborhoods: Index of Perceptions of Neighborhood Safety
Description: as for outcome 131
Time Frame: Age 24 months
Reporting Status: Not Posted

133. Secondary Outcome: Housing and Neighborhoods: Index of Perceptions of Neighborhood Safety
Description: Index of Perceptions of Neighborhood Safety measured by an additive index of survey items (see Appendix Table 8 in "Analysis Plan and Measures" document for items).
  Minimum score: 0; Maximum score: 6. Higher score indicates a better outcome.
  We will estimate the statistical significance of the entire family of related measures in the Housing and Neighborhoods outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Kling, J.R., Liebman, J.B., Katz, L.F. (2007). Experimental analysis of neighborhood effects. Econometrica, 75(1), 83-119.
Time Frame: Age 36 months
Reporting Status: Not Posted

134. Secondary Outcome: Housing and Neighborhoods: Index of Housing Quality
Description: Index of Housing Quality measured by an additive index of survey items(see Appendix Table 8 in "Analysis Plan and Measures" document for items).
  We will estimate the statistical significance of the entire family of related measures in the Housing and Neighborhoods outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Kling, J.R., Liebman, J.B., Katz, L.F. (2007). Experimental analysis of neighborhood effects. Econometrica, 75(1), 83-119.
Time Frame: Age 12 months
Reporting Status: Not Posted

135. Secondary Outcome: Housing and Neighborhoods: Index of Housing Quality
Description: Index of Housing Quality measured by an additive index of survey items (see Appendix Table 8 in "Analysis Plan and Measures" document for items).
  We will estimate the statistical significance of the entire family of related measures in the Housing and Neighborhoods outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Kling, J.R., Liebman, J.B., Katz, L.F. (2007). Experimental analysis of neighborhood effects. Econometrica, 75(1), 83-119.
Time Frame: Age 24 months
Reporting Status: Not Posted

136. Secondary Outcome: Housing and Neighborhoods: Excessive Residential Mobility
Description: Excessive Residential Mobility measured by survey items (see Appendix Table 8 in "Analysis Plan and Measures" document for items).
  We will estimate the statistical significance of the entire family of related measures in the Housing and Neighborhoods outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Kling, J.R., Liebman, J.B., Katz, L.F. (2007). Experimental analysis of neighborhood effects. Econometrica, 75(1), 83-119.
Time Frame: Age 12 months
Reporting Status: Not Posted

137. Secondary Outcome: Housing and Neighborhoods: Excessive Residential Mobility
Description: as for outcome 136
Time Frame: Age 24 months
Reporting Status: Not Posted

138. Secondary Outcome: Housing and Neighborhoods: Excessive Residential Mobility
Description: Excessive Residential Mobility measured by survey items (see Appendix Table 8 in "Analysis Plan and Measures" document for items).
  Minimum score: 0; Maximum score: 1. Higher score indicates worse outcome.
  We will estimate the statistical significance of the entire family of related measures in the Housing and Neighborhoods outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Kling, J.R., Liebman, J.B., Katz, L.F. (2007). Experimental analysis of neighborhood effects. Econometrica, 75(1), 83-119.
Time Frame: Age 36 months
Reporting Status: Not Posted

139. Secondary Outcome: Housing and Neighborhoods: Homelessness
Description: Homelessness measured by survey items (see Appendix Table 8 in "Analysis Plan and Measures" document for items).
  We will estimate the statistical significance of the entire family of related measures in the Housing and Neighborhoods outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Kling, J.R., Liebman, J.B., Katz, L.F. (2007). Experimental analysis of neighborhood effects. Econometrica, 75(1), 83-119.
Time Frame: Age 12 months
Reporting Status: Not Posted

140. Secondary Outcome: Housing and Neighborhoods: Homelessness
Description: as for outcome 139
Time Frame: Age 24 months
Reporting Status: Not Posted

141. Secondary Outcome: Housing and Neighborhoods: Homelessness
Description: Homelessness measured by survey items (see Appendix Table 8 in "Analysis Plan and Measures" document for items).
  Minimum score: 0; Maximum score: 1. Higher score indicates worse outcome.
  We will estimate the statistical significance of the entire family of related measures in the Housing and Neighborhoods outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Kling, J.R., Liebman, J.B., Katz, L.F. (2007). Experimental analysis of neighborhood effects. Econometrica, 75(1), 83-119.
Time Frame: Age 36 months
Reporting Status: Not Posted

142. Secondary Outcome: Housing and Neighborhoods: Neighborhood Poverty
Description: Neighborhood Poverty measured by the proportion of residents in the respondent's census tract that are below the poverty line, using census data.
  We will estimate the statistical significance of the entire family of related measures in the Housing and Neighborhoods outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Kling, J.R., Liebman, J.B., Katz, L.F. (2007). Experimental analysis of neighborhood effects. Econometrica, 75(1), 83-119.
Time Frame: Age 12 months
Reporting Status: Not Posted

143. Secondary Outcome: Housing and Neighborhoods: Neighborhood Poverty
Description: as for outcome 142
Time Frame: Age 24 months
Reporting Status: Not Posted

144. Secondary Outcome: Housing and Neighborhoods: Neighborhood Poverty
Description: as for outcome 142
Time Frame: Age 36 months
Reporting Status: Not Posted

145. Secondary Outcome: Housing and Neighborhoods: Neighborhood Poverty
Description: as for outcome 142
Time Frame: Age 48 months
Reporting Status: Not Posted

146. Secondary Outcome: Housing and Neighborhoods: Neighborhood Poverty
Description: Neighborhood Poverty measured by the proportion of residents in the respondent's census tract that are below the poverty line, using census data. Expect less neighborhood poverty in the high-cash group.
  Reference:
  Kling, J.R., Liebman, J.B., Katz, L.F. (2007). Experimental analysis of neighborhood effects. Econometrica, 75(1), 83-119.
Time Frame: Age 6
Reporting Status: Not Posted

147. Secondary Outcome: Housing and Neighborhoods: Neighborhood Poverty
Description: as for outcome 146
Time Frame: Age 8
Reporting Status: Not Posted

148. Secondary Outcome: Family and Maternal Perceived Stress: Perceived Stress
Description: Perceived Stress measured by the Perceived Stress Scale (PSS).
  We will estimate the statistical significance of the entire family of related measures in the Family and Maternal Perceived Stress outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Cohen, S., Kamarck, T., & Mermelstein, R. (1994). Perceived stress scale. Measuring stress: A guide for health and social scientists.
Time Frame: Age 12 months
Reporting Status: Not Posted

149. Secondary Outcome: Family and Maternal Perceived Stress: Parenting Stress
Description: Parenting Stress measured by the Aggravation in Parenting Scale.
  We will estimate the statistical significance of the entire family of related measures in the Family and Maternal Perceived Stress outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  The Child Development Supplement to the Panel Study of Income Dynamics, retrieved from https://psidonline.isr.umich.edu/cds/cdsi_usergd.pdf
Time Frame: Age 12 months
Reporting Status: Not Posted

150. Secondary Outcome: Family and Maternal Perceived Stress: Perceived Stress
Description: as for outcome 148
Time Frame: Age 24 months
Reporting Status: Not Posted

151. Secondary Outcome: Family and Maternal Perceived Stress: Parenting Stress
Description: as for outcome 149
Time Frame: Age 24 months
Reporting Status: Not Posted

152. Secondary Outcome: Family and Maternal Perceived Stress: Perceived Stress
Description: Perceived Stress measured by the Perceived Stress Scale (PSS).
  Minimum score: 0; Maximum score: 32. Higher score indicates worse outcome.
  We will estimate the statistical significance of the entire family of related measures in the Family and Maternal Perceived Stress outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Cohen, S., Kamarck, T., & Mermelstein, R. (1994). Perceived stress scale. Measuring stress: A guide for health and social scientists.
Time Frame: Age 36 months
Reporting Status: Not Posted

153. Secondary Outcome: Family and Maternal Perceived Stress: Parenting Stress
Description: Parenting Stress measured by the Aggravation in Parenting Scale.
  Note: Index dropped from age 4 survey owing to time constraints
  Reference:
  The Child Development Supplement to the Panel Study of Income Dynamics, retrieved from https://psidonline.isr.umich.edu/cds/cdsi_usergd.pdf
Time Frame: Age 48 months
Reporting Status: Not Posted

154. Secondary Outcome: Maternal Happiness and Optimism: Global Happiness
Description: Global Happiness measured by survey item (see Appendix Table 8 in "Analysis Plan and Measures" document for items).
  We will estimate the statistical significance of the entire family of related measures in the Maternal Happiness and Optimism outcome cluster using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  The General Social Survey from NORC at the University of Chicago, retrieved from: http://gss.norc.org/Get-Documentation/questionnaires
Time Frame: Age 12 months
Reporting Status: Not Posted

155. Secondary Outcome: Maternal Happiness and Optimism: Global Happiness
Description: as for outcome 154
Time Frame: Age 24 months
Reporting Status: Not Posted

156. Secondary Outcome: Maternal Happiness and Optimism: Global Happiness
Description: Global Happiness measured by survey item (see Appendix Table 8 in "Analysis Plan and Measures" document for items).
  Minimum score: 1; Maximum score: 3. Higher score indicates better outcome.
  We will estimate the statistical significance of the entire family of related measures in the Maternal Happiness and Optimism outcome cluster using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  The General Social Survey from NORC at the University of Chicago, retrieved from: http://gss.norc.org/Get-Documentation/questionnaires
Time Frame: Age 36 months
Reporting Status: Not Posted

157. Secondary Outcome: Maternal Happiness
Description: Global Happiness measured by survey item (see Appendix Table 10 in "Analysis Plan and Measures" document for items).
  Minimum score: 1; Maximum score: 3. Higher score indicates better outcome. Expect higher score in high-cash group.
  We will estimate the statistical significance of the entire family of related measures in the Maternal Happiness and Optimism outcome cluster using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  The General Social Survey from NORC at the University of Chicago, retrieved from: http://gss.norc.org/Get-Documentation/questionnaires
Time Frame: Age 6
Reporting Status: Not Posted

158. Secondary Outcome: Maternal Happiness
Description: as for outcome 157
Time Frame: Age 8
Reporting Status: Not Posted

159. Secondary Outcome: Maternal Happiness and Optimism: Optimism
Description: Optimism measured by the Adult Hope Scale.
  We will estimate the statistical significance of the entire family of related measures in the Maternal Happiness and Optimism outcome cluster using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Snyder, C.R., Harris, C., Anderson, J.R., Holleran, S.A., Irving, L.M., Sigmon, S.T., Yoshinobu, L., Gibb, J., Langelle, C., Harney, P. (1991). The will and the ways: development and validation of an individual-differences measure of hope. Journal of Personality and Social Psychology, 60(4), 570-585.
Time Frame: Age 12 months
Reporting Status: Not Posted

160. Secondary Outcome: Maternal Happiness and Optimism: Optimism
Description: as for outcome 159
Time Frame: Age 24 months
Reporting Status: Not Posted

161. Secondary Outcome: Maternal Happiness and Optimism: Optimism
Description: Optimism measured by the Adult Hope Scale.
  Minimum score: 10; Maximum score: 30. Higher score indicates better outcome.
  We will estimate the statistical significance of the entire family of related measures in the Maternal Happiness and Optimism outcome cluster using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Snyder, C.R., Harris, C., Anderson, J.R., Holleran, S.A., Irving, L.M., Sigmon, S.T., Yoshinobu, L., Gibb, J., Langelle, C., Harney, P. (1991). The will and the ways: development and validation of an individual-differences measure of hope. Journal of Personality and Social Psychology, 60(4), 570-585.
Time Frame: Age 36 months
Reporting Status: Not Posted

162. Secondary Outcome: Maternal Physiological Stress: Maternal Hair Cortisol
Description: Measured by maternal hair cortisol.
  Reference:
  Ursache, A., Merz, E.C., Melvin, S., Meyer, J., Noble, K.G. (2017). Socioeconomic status, hair cortisol and internalizing symptoms in parents and children. Psychoneuroendocrinology, 78, 142-150.
Time Frame: Age 12 months
Reporting Status: Not Posted

163. Secondary Outcome: Maternal Physiological Stress: Maternal Hair Cortisol
Description: Measured by maternal hair cortisol.
  Note: Our original plan was to measure physiological stress using hair cortisol concentration. The first several months of data collection revealed large racial and ethnic differences in willingness to provide a hair sample, due to both cultural and practical reasons. Because of the large amounts of non-random missing data, which would both compromise our statistical power and limit the generalizability of any findings, we dropped hair cortisol from our data collection procedures on October 25, 2022.
  Reference:
  Ursache, A., Merz, E.C., Melvin, S., Meyer, J., Noble, K.G. (2017). Socioeconomic status, hair cortisol and internalizing symptoms in parents and children. Psychoneuroendocrinology, 78, 142-150.
Time Frame: Age 48 months
Reporting Status: Not Posted

164. Secondary Outcome: Maternal Executive Function
Description: Measured by the Minnesota Executive Function Scale.
  Minimum score: 60; Maximum score: 140. Higher score indicates a better outcome.
  Reference:
  Carlson, S. M., & Zelazo, P. D. (2014). Minnesota Executive Function Scale: Test Manual. St. Paul, MN: Reflection Sciences, Inc.
  Carlson, S. M. (2017). Minnesota Executive Function Scale: Technical Report, v. 2. St. Paul, MN: Reflection Sciences, Inc.
Time Frame: Age 48 months
Reporting Status: Not Posted

165. Secondary Outcome: Maternal Executive Function
Description: Measured by the Minnesota Executive Function Scale (MEFS) Minimum score: 60; Maximum score: 140. Higher score indicates a better outcome. We expect a higher value of the maternal MEFS standardized score for the high-cash gift group mothers than the low-cash gift mothers.
  Reference:
  Carlson, S. M., & Zelazo, P. D. (2014). Minnesota Executive Function Scale: Test Manual. St. Paul, MN: Reflection Sciences, Inc.
  Carlson, S. M. (2017). Minnesota Executive Function Scale: Technical Report, v. 2. St. Paul, MN: Reflection Sciences, Inc.
  Reflection Sciences (2021). Minnesota executive function scale technical report. Reflection Sciences. https://reflectionsciences.com/wp-content/uploads/MEFS-Technical-Report-July-2021.pdf
Time Frame: Age 6
Reporting Status: Not Posted

166. Secondary Outcome: Maternal Executive Function
Description: Measured by the Minnesota Executive Function Scale (MEFS). Minimum score: 60; Maximum score: 140. Higher score indicates a better outcome. We expect a higher value of the maternal MEFS standardized score for the high-cash gift group mothers than the low-cash gift mothers.
  Reference:
  Carlson, S. M., & Zelazo, P. D. (2014). Minnesota Executive Function Scale: Test Manual. St. Paul, MN: Reflection Sciences, Inc.
  Carlson, S. M. (2017). Minnesota Executive Function Scale: Technical Report, v. 2. St. Paul, MN: Reflection Sciences, Inc.
  Reflection Sciences (2021). Minnesota executive function scale technical report. Reflection Sciences. https://reflectionsciences.com/wp-content/uploads/MEFS-Technical-Report-July-2021.pdf
Time Frame: Age 8
Reporting Status: Not Posted

167. Secondary Outcome: Maternal Mental Health: Index of Maternal Depression
Description: Index of Maternal Depression measured by the Patient Health Questionnaire (PHQ-8).
  Min value: 0; Max value: 24
  Higher score indicates worse outcome.
  We will estimate the statistical significance of the entire family of related measures in the Maternal Mental Health outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Kroenke, K. & Spitzer, R.L. (2002). The PHQ-9: a new depression diagnostic and severity measure. Psychiatric annals, 32(9), 509-515.
Time Frame: Age 12 months
Reporting Status: Not Posted

168. Secondary Outcome: Maternal Mental Health: Index of Maternal Depression
Description: as for outcome 167
Time Frame: Age 24 months
Reporting Status: Not Posted

169. Secondary Outcome: Maternal Mental Health: Index of Maternal Depression
Description: Index of Maternal Depression measured by the Patient Health Questionnaire (PHQ-8).
  Min value: 0; Max value: 24. Higher score indicates worse outcome.
  We will estimate the statistical significance of the entire family of related measures in the Maternal Mental Health outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Kroenke, K. & Spitzer, R.L. (2002). The PHQ-9: a new depression diagnostic and severity measure. Psychiatric annals, 32(9), 509-515.
Time Frame: Age 36 months
Reporting Status: Not Posted

170. Secondary Outcome: Maternal Mental Health: Index of Maternal Depression
Description: as for outcome 169
Time Frame: Age 48 months
Reporting Status: Not Posted

171. Secondary Outcome: Maternal Mental Health: Index of Maternal Depression
Description: Index of Maternal Depression measured by the Patient Health Questionnaire (PHQ-8).
  Min value: 0; Max value: 24. Higher score indicates worse outcome. We expect less depression in the high- as opposed to low-cash group.
  We will estimate the statistical significance of the entire family of related measures in the Maternal Mental Health outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Kroenke, K. & Spitzer, R.L. (2002). The PHQ-9: a new depression diagnostic and severity measure. Psychiatric annals, 32(9), 509-515.
Time Frame: Age 6
Reporting Status: Not Posted

172. Secondary Outcome: Maternal Mental Health: Index of Maternal Depression
Description: as for outcome 171
Time Frame: Age 8
Reporting Status: Not Posted

173. Secondary Outcome: Maternal Mental Health: Index of Maternal Anxiety
Description: Index of Maternal Anxiety measured by the Beck Anxiety Inventory.
  We will estimate the statistical significance of the entire family of related measures in the Maternal Mental Health outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Steer, R.A. & Beck, A.T., (1997). Beck Anxiety Inventory. In C.P. Zalaquett & R.J. Wood (Eds), Evaluating stress: A book of resources (pp. 23-40). Lanham, MD, US: Scarecrow Education
Time Frame: Age 12 months
Reporting Status: Not Posted

174. Secondary Outcome: Maternal Mental Health: Index of Maternal Anxiety
Description: Index of Maternal Anxiety measured by the GAD-7.
  We will estimate the statistical significance of the entire family of related measures in the Maternal Mental Health outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Spitzer RL, Kroenke K, Williams JBW, Löwe B. A Brief Measure for Assessing Generalized Anxiety Disorder: The GAD-7. Arch Intern Med. 2006;166(10):1092-1097. doi:10.1001/archinte.166.10.1092
Time Frame: Age 24 months
Reporting Status: Not Posted

175. Secondary Outcome: Maternal Mental Health: Index 1 of Maternal Anxiety
Description: as for outcome 174
Time Frame: Age 36 months
Reporting Status: Not Posted

176. Secondary Outcome: Maternal Mental Health: Index 2 of Maternal Anxiety
Description: Index of Maternal Anxiety measured by the Beck Anxiety Inventory.
  Min value: 0; Max value: 44. Higher score indicates worse outcome.
  We will estimate the statistical significance of the entire family of related measures in the Maternal Mental Health outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Steer, R.A. & Beck, A.T., (1997). Beck Anxiety Inventory. In C.P. Zalaquett & R.J. Wood (Eds), Evaluating stress: A book of resources (pp. 23-40). Lanham, MD, US: Scarecrow Education
Time Frame: Age 36 months
Reporting Status: Not Posted

177. Secondary Outcome: Maternal Mental Health: Index of Maternal Anxiety
Description: as for outcome 174
Time Frame: Age 48 months
Reporting Status: Not Posted

178. Secondary Outcome: Maternal Mental Health: Index of Maternal Anxiety
Description: Index of Maternal Anxiety measured by the GAD-7. Min value: 0; Max value: 21. Higher score indicates worse outcome. We expect less anxiety in the high- as opposed to low-cash group.
  We will estimate the statistical significance of the entire family of related measures in the Maternal Mental Health outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Spitzer RL, Kroenke K, Williams JBW, Löwe B. A Brief Measure for Assessing Generalized Anxiety Disorder: The GAD-7. Arch Intern Med. 2006;166(10):1092-1097. doi:10.1001/archinte.166.10.1092
Time Frame: Age 6
Reporting Status: Not Posted

179. Secondary Outcome: Maternal Mental Health: Index of Maternal Anxiety
Description: as for outcome 178
Time Frame: Age 8
Reporting Status: Not Posted

180. Secondary Outcome: Maternal Substance Abuse: Alcohol and Cigarette Use
Description: Alcohol and Cigarette Use measured by an additive index of survey items (see Appendix Table 8 in "Analysis Plan and Measures" document for items).
  We will estimate the statistical significance of the entire family of related measures in the Maternal Substance Abuse outcome cluster using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Kling, J.R., Liebman, J.B., Katz, L.F. (2007). Experimental analysis of neighborhood effects. Econometrica, 75(1), 83-119.
Time Frame: Age 12 months
Reporting Status: Not Posted

181. Secondary Outcome: Maternal Substance Abuse: Alcohol and Cigarette Use
Description: Alcohol and Cigarette Use measured by an additive index of survey items (see Appendix Table 8 in "Analysis Plan and Measures" document for items).
  Minimum score: 0; Maximum score: 8. Higher score indicates worse outcome.
  We will estimate the statistical significance of the entire family of related measures in the Maternal Substance Abuse outcome cluster using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Kling, J.R., Liebman, J.B., Katz, L.F. (2007). Experimental analysis of neighborhood effects. Econometrica, 75(1), 83-119.
Time Frame: Age 36 months
Reporting Status: Not Posted

182. Secondary Outcome: Maternal Substance Abuse: Opioid Use
Description: Opioid Use measured by a survey item (see Appendix Table 8 in "Analysis Plan and Measures" document for item).
  We will estimate the statistical significance of the entire family of related measures in the Maternal Substance Abuse outcome cluster using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Kling, J.R., Liebman, J.B., Katz, L.F. (2007). Experimental analysis of neighborhood effects. Econometrica, 75(1), 83-119.
Time Frame: Age 12 months
Reporting Status: Not Posted

183. Secondary Outcome: Maternal Substance Abuse: Opioid Use
Description: Opioid Use measured by a survey item (see Appendix Table 8 in "Analysis Plan and Measures" document for item).
  Minimum score: 0; Maximum score: 4. Higher score indicates worse outcome.
  We will estimate the statistical significance of the entire family of related measures in the Maternal Substance Abuse outcome cluster using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Kling, J.R., Liebman, J.B., Katz, L.F. (2007). Experimental analysis of neighborhood effects. Econometrica, 75(1), 83-119.
Time Frame: Age 36 months
Reporting Status: Not Posted

184. Secondary Outcome: Chaos in the Home: Index of Chaos in the Home
Description: Measured by the Home Environment Chaos Scale.
  Reference:
  Evans, G.W., Gonnella, C., Marcynyszyn, L.A., Gentile, L, & Salpekar, N. (2005). The role of chaos in poverty and children's socioemotional adjustment. Psychological Science, 16(7), 560-565.
Time Frame: Age 12 months
Reporting Status: Not Posted

185. Secondary Outcome: Chaos in the Home: Index of Chaos in the Home
Description: as for outcome 184
Time Frame: Age 24 months
Reporting Status: Not Posted

186. Secondary Outcome: Maternal Relationships: Physical Abuse
Description: Measured by a survey item (see Appendix Table 8 in "Analysis Plan and Measures" document for item).
  We will estimate the statistical significance of the entire family of related measures in the Maternal Relationships outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  User's Guide for the Fragile Families and Child Wellbeing Study Public Data, Year 3. (2018). Retrieved from: https://fragilefamilies.princeton.edu/sites/fragilefamilies/files/year_3_guide.pdf
Time Frame: Age 12 months
Reporting Status: Not Posted

187. Secondary Outcome: Maternal Relationships: Physical Abuse
Description: as for outcome 186
Time Frame: Age 24 months
Reporting Status: Not Posted

188. Secondary Outcome: Maternal Relationships: Frequency of Arguing
Description: as for outcome 186
Time Frame: Age 12 months
Reporting Status: Not Posted

189. Secondary Outcome: Maternal Relationships: Frequency of Arguing
Description: as for outcome 186
Time Frame: Age 24 months
Reporting Status: Not Posted

190. Secondary Outcome: Maternal Relationships: Relationship Quality
Description: Measured by an additive index of survey items (see Appendix Table 8 in "Analysis Plan and Measures" document for items).
  We will estimate the statistical significance of the entire family of related measures in the Maternal Relationships outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  User's Guide for the Fragile Families and Child Wellbeing Study Public Data, Year 3. (2018). Retrieved from: https://fragilefamilies.princeton.edu/sites/fragilefamilies/files/year_3_guide.pdf
Time Frame: Age 12 months
Reporting Status: Not Posted

191. Secondary Outcome: Maternal Relationships: Relationship Quality
Description: Measured by a dichotomous indicator generated from an additive index of survey items (see Appendix Table 8 in "Analysis Plan and Measures" document for items and cutoff point for high or low quality).
  We will estimate the statistical significance of the entire family of related measures in the Maternal Relationships outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  User's Guide for the Fragile Families and Child Wellbeing Study Public Data, Year 3. (2018). Retrieved from: https://fragilefamilies.princeton.edu/sites/fragilefamilies/files/year_3_guide.pdf
Time Frame: Age 24 months
Reporting Status: Not Posted

192. Secondary Outcome: Maternal Relationships: Relationship Quality
Description: Measured by a dichotomous indicator generated from an additive index of survey items (see Appendix Table 8 in "Analysis Plan and Measures" document for items and cutoff point for high or low quality).
  Minimum score: 0; Maximum score: 1. Higher score indicates worse outcome.
  We will estimate the statistical significance of the entire family of related measures in the Maternal Relationships outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  User's Guide for the Fragile Families and Child Wellbeing Study Public Data, Year 3. (2018). Retrieved from: https://fragilefamilies.princeton.edu/sites/fragilefamilies/files/year_3_guide.pdf
Time Frame: Age 36 months
Reporting Status: Not Posted

193. Secondary Outcome: Maternal Physical Health: Global Health
Description: Global Health measured by one survey item (see Appendix Table 8 in "Analysis Plan and Measures" document for items).
  We will estimate the statistical significance of the entire family of related measures in the Maternal Physical Health outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Idler, E. L., & Benyamini, Y. (1997). Self-rated health and mortality: a review of twenty-seven community studies. Journal of health and social behavior, 21-37.
Time Frame: Age 12 months
Reporting Status: Not Posted

194. Secondary Outcome: Maternal Physical Health: Global Health
Description: Global Health measured by one survey item (see Appendix Table 8 in "Analysis Plan and Measures" document for items).
  We will estimate the statistical significance of the entire family of related measures in the Maternal Physical Health outcome measured during the same wave cluster using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Idler, E. L., & Benyamini, Y. (1997). Self-rated health and mortality: a review of twenty-seven community studies. Journal of health and social behavior, 21-37.
Time Frame: Age 24 months
Reporting Status: Not Posted

195. Secondary Outcome: Maternal Physical Health: Global Health
Description: Global Health measured by one survey item (see Appendix Table 10 in "Analysis Plan and Measures" document for items). Expect better health for high-cash group.
  We will estimate the statistical significance of the entire family of related measures in the Maternal Physical Health outcome measured during the same wave cluster using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Idler, E. L., & Benyamini, Y. (1997). Self-rated health and mortality: a review of twenty-seven community studies. Journal of health and social behavior, 21-37.
Time Frame: Age 6
Reporting Status: Not Posted

196. Secondary Outcome: Maternal Physical Health: Global Health
Description: as for outcome 195
Time Frame: Age 8
Reporting Status: Not Posted

197. Secondary Outcome: Maternal Physical Health: Sleep
Description: Sleep measured by an additive index of survey items (see Appendix Table 8 in "Analysis Plan and Measures" document for items).
  Minimum score: 4; Maximum score: 20. Higher score indicates a better outcome.
  We will estimate the statistical significance of the entire family of related measures in the Maternal Physical Health outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Kling, J.R., Liebman, J.B., Katz, L.F. (2007). Experimental analysis of neighborhood effects. Econometrica, 75(1), 83-119.
Time Frame: Age 12 months
Reporting Status: Not Posted

198. Secondary Outcome: Maternal Physical Health: Sleep
Description: Sleep measured by an additive index of survey items (see Appendix Table 8 in "Analysis Plan and Measures" document for items).
  Minimum score: 3; Maximum score: 15. Higher score indicates a better outcome.
  We will estimate the statistical significance of the entire family of related measures in the Maternal Physical Health outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Kling, J.R., Liebman, J.B., Katz, L.F. (2007). Experimental analysis of neighborhood effects. Econometrica, 75(1), 83-119.
Time Frame: Age 36 months
Reporting Status: Not Posted

199. Secondary Outcome: Maternal Physical Health: Body Mass Index
Description: Body Mass Index measured by Center for Disease Control and Prevention (CDC) growth charts.
  Reference:
  Kuczmarski, R. J. (2000). CDC growth charts; United States.
Time Frame: Age 48 months
Reporting Status: Not Posted

200. Secondary Outcome: Maternal Physical Health: Body Mass Index
Description: Body Mass Index measured by Center for Disease Control and Prevention (CDC) growth charts.
  Dichotomous measure based on CDC BMI percentile scales We expect to see a reduced percentage of overweight or obese (BMI greater than or equal to 25) mothers in the high-cash gift group compared to the low-cash gift group. We will report mean BMI of the two groups in descriptive analyses.
  Reference:
  Kuczmarski, R. J. (2000). CDC growth charts; United States.
Time Frame: Age 6
Reporting Status: Not Posted

201. Secondary Outcome: Maternal Physical Health: Body Mass Index
Description: as for outcome 200
Time Frame: Age 8
Reporting Status: Not Posted

202. Secondary Outcome: Parent-Child Interaction Quality: Adult Word Count
Description: Adult Word Count measured by LENA Processing Software.
  We will estimate the statistical significance of the entire family of related measures in the Parent-Child Interaction Quality outcome cluster using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Xu, D., Yapanel, U., & Gray, S. (2009). Reliability of the LENA Language Environment Analysis System in young children's natural home environment. LENA Foundation.
Time Frame: Age 12 months
Reporting Status: Not Posted

203. Secondary Outcome: Parent-Child Interaction Quality: Conversational Turns
Description: Conversational Turns measured by LENA Processing Software.
  We will estimate the statistical significance of the entire family of related measures in the Parent-Child Interaction Quality outcome cluster using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Xu, D., Yapanel, U., & Gray, S. (2009). Reliability of the LENA Language Environment Analysis System in young children's natural home environment. LENA Foundation.
Time Frame: Age 12 months
Reporting Status: Not Posted

204. Secondary Outcome: Parent-Child Interaction Quality: Index of Mother's Positive Parenting Behaviors
Description: Measured using PICCOLO coding of parenting behaviors from the total of four sub-scales (affection, responsiveness, encouragement and teaching) with responses ranging from 0: absent, 1: barely, 2: clearly. Parent child interaction task and script adapted from the NICHD Study of Early Child Care and Youth Development.
  We will estimate the statistical significance of the entire family of related measures in the Parent-Child Interaction Quality outcome cluster using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Roggman, et al. (2013). Observations Linked to Outcomes (PICCOLO) Of Diverse Ethnic Groups. Infant Mental Health Journal, 34(4), 290-306.
  Griffin, J. A., & Friedman, S. L. (2007). NICHD Study of Early Childcare and Youth Development. National Institute of Health
  Belsky, J., et al. (2007). Are there long-term effects of early child care?. Child development, 78(2), 681-701.
Time Frame: Age 12 months
Reporting Status: Not Posted

205. Secondary Outcome: Parent-Child Interaction Quality: Index of Mother's Positive Parenting Behaviors
Description: Measured using PICCOLO coding of parenting behaviors from the total of four sub-scales (affection, responsiveness, encouragement and teaching) with responses ranging from 0: absent, 1: barely, 2: clearly. Parent child interaction task and script adapted from the NICHD Study of Early Child Care and Youth Development.
  Reference:
  Roggman, et al. (2013). Observations Linked to Outcomes (PICCOLO) Of Diverse Ethnic Groups. Infant Mental Health Journal, 34(4), 290-306.
  Griffin, J. A., & Friedman, S. L. (2007). NICHD Study of Early Childcare and Youth Development. National Institute of Health
  Belsky, J., et al. (2007). Are there long-term effects of early child care?. Child development, 78(2), 681-701.
Time Frame: Age 48 months
Reporting Status: Not Posted

206. Secondary Outcome: Parent-Child Interaction Quality: Index of Mother's Positive Parenting Behaviors
Description: Block play and grocery shopping game. Grocery shopping game task and script adapted from Leyva et al., 2017 and Leyva et al., 2019. Coding: Measured using Emotional Availability scale (EAS) - 4th Edition middle childhood/youth version (Biringen et al., 2008; Biringen et al., 2014) coding of parenting behaviors from a total of four maternal sub-scales (sensitivity, structuring, non-intrusiveness, and non-hostility) with responses scored on a 7-point scale across the two PCI tasks. The additive total composite score will be pre-registered. We hypothesize a higher composite score for the high-cash gift group relative to the low-cash gift group. Please see details of confirmatory factor analysis, exploratory analysis, and all references in Table 10 in the Statistical Analysis Plan.
Time Frame: Age 6
Reporting Status: Not Posted

207. Secondary Outcome: Parent-Child Interaction Quality: Index of Mother's Positive Parenting Behaviors
Description: Two tasks to be determined. Coding: Measured using Emotional Availability scale (EAS) - 4th Edition middle childhood/youth version (Biringen et al., 2008; Biringen et al., 2014) coding of parenting behaviors from a total of four maternal sub-scales (sensitivity, structuring, non-intrusiveness, and non-hostility) with responses scored on a 7-point scale across the two PCI tasks. The additive total composite score will be pre-registered. We hypothesize a higher composite score for the high-cash gift group relative to the low-cash gift group. Please see details of confirmatory factor analysis, exploratory analysis, and all references in Table 10 in the Statistical Analysis Plan.
Time Frame: Age 8
Reporting Status: Not Posted

208. Secondary Outcome: Parent-Child Interaction Quality: Maternal Language Quantity
Description: Measured by the total number of word tokens (adult word count) in maternal speech during the parent-child interaction tasks (Anderson et al 2021; Rowe, 2008; Rowe, 2012). Coded through transcripts at the utterance level. We hypothesize a higher adult word count for mothers in the high-cash gift group relative to the low-cash gift group.
  References:
  Anderson, N. J., Graham, S. A., Prime, H., Jenkins, J. M., & Madigan, S. (2021). Linking quality and quantity of parental linguistic input to child language skills: A meta-analysis. Child Development, 92(2), 484-501.
  Rowe, M. (2008). Child-directed speech: relation to socioeconomic status, knowledge of child development and child vocabulary skill. Journal of Child Language, 35, 185-205. doi:10.1017/S0305000907008343 Rowe, M. (2012). A Longitudinal Investigation of the Role of Quantity and Quality of Child-Directed Speech in Vocabulary Development. Child Development, 83(5), 1762-1774.
Time Frame: Age 6
Reporting Status: Not Posted

209. Secondary Outcome: Parent-Child Interaction Quality: Maternal Language Quantity
Description: as for outcome 208
Time Frame: Age 8
Reporting Status: Not Posted

210. Secondary Outcome: Parent-Child Interaction Quality: Maternal Language Quality
Description: Measured through three indicators of quality: Mean length of utterance (MLU; average number of morphemes per utterance), word types (number of different word roots produced) as indicators of language complexity and diversity, respectively (Anderson et al 2021; Rowe, 2008; Rowe, 2012), and the proportion of utterances that are wh- questions -What, Where, When, Which, Why, Who, and How (referential and inferential questions)-(Luo et al., 2022; Cristofaro & Tamis-LeMonda, 2012) in maternal speech during the parent-child interaction tasks. Language quality variables will be coded through transcripts at the utterance level. We hypothesize higher language quality scores, either the composite factor or the individual scores, for the high-cash gift group relative to the low-cash gift group. Please see details of planned analysis and all references in Table 10 in the Statistical Analysis Plan.
Time Frame: Age 6
Reporting Status: Not Posted

211. Secondary Outcome: Parent-Child Interaction Quality: Maternal Language Quality
Description: as for outcome 210
Time Frame: Age 8
Reporting Status: Not Posted

212. Secondary Outcome: Maternal Epigenetic Pace of Aging
Description: Measured using method reported in Appendix Table 8 in "Analysis Plan and Measures" document. Please also see preregistration at OSF: https://osf.io/ahv2p/?view_only=
  Reference:
  Belsky, W. D. et al. (2020). Quantification of the pace of biological aging in humans through blood test, the DunedinPoAm DNA methylation algorithm. eLife 9:e54870. https://doi.org/10.7554/eLife.54870
  Belsky, W. D. et al. (2022). DunedinPACE, a DNA methylation biomarker of the pace of aging. eLife 11:e73420. https://doi.org/10.7554/eLife.73420
Time Frame: Age 48 months
Reporting Status: Not Posted

213. Secondary Outcome: Maternal Epigenetic Pace of Aging
Description: Expect slower DunedinPACE- pace of aging in high-cash group: Methylation pace of aging was developed from DNA-methylation analysis of Pace of Aging in the Dunedin Study birth cohort (Belsky et al., 2022).. Pace of Aging is a composite phenotype derived from analysis of longitudinal change in 18 biomarkers of organ-system integrity (Belsky et al., 2015). Increments of methylation pace of aging correspond to "years" of physiological change occurring per 12-months of chronological time. We will also report GrimAge Acceleration and PhenoAge Acceleration as exploratory analyses. GrimAge represents a DNA-methylation metric designed to predict morbidity and mortality (Lu et al., 2019). Please see details and references in Appendix Table 10.
Time Frame: Age 6
Reporting Status: Not Posted

214. Secondary Outcome: Maternal Epigenetic Pace of Aging
Description: as for outcome 213
Time Frame: Age 8
Reporting Status: Not Posted

215. Secondary Outcome: Maternal DNA Methylation
Description: Measured using method reported in Appendix Table 8 in "Analysis Plan and Measures" document. Please also see preregistration at OSF: https://osf.io/ahv2p/?view_only=
  Reference:
  McCartney, D.L., Hillary, R.F., Conole, E.L.S. et al. Blood-based epigenome-wide analyses of cognitive abilities. Genome Biol 23, 26 (2022). https://doi.org/10.1186/s13059-021-02596-5
Time Frame: Age 48 months
Reporting Status: Not Posted

216. Secondary Outcome: Frequency of Parent-Child Activity: Self-Report of Parent-Child Activities
Description: Frequency of Parent-Child Activity measured by an additive index of survey items (see Appendix Table 8 in "Analysis Plan and Measures" document for items).
  Reference:
  Rodriguez, E. T., & Tamis-LeMonda, C. S. (2011). Trajectories of the home learning environment across the first 5 years: Associations with children's vocabulary and literacy skills at prekindergarten. Child development, 82(4), 1058-1075.
Time Frame: Age 12 months
Reporting Status: Not Posted

217. Secondary Outcome: Frequency of Parent-Child Activity: Self-Report of Parent-Child Activities
Description: as for outcome 216
Time Frame: Age 24 months
Reporting Status: Not Posted

218. Secondary Outcome: Frequency of Parent-Child Activity: Self-Report of Parent-Child Activities
Description: Frequency of Parent-Child Activity measured by an additive index of survey items (see Appendix Table 8 in "Analysis Plan and Measures" document for items).
  Minimum score: 4; Maximum score: 20. Higher score indicates better outcome.
  Reference:
  Rodriguez, E. T., & Tamis-LeMonda, C. S. (2011). Trajectories of the home learning environment across the first 5 years: Associations with children's vocabulary and literacy skills at prekindergarten. Child development, 82(4), 1058-1075.
Time Frame: Age 36 months
Reporting Status: Not Posted

219. Secondary Outcome: Frequency of Parent-Child Activity: Self-Report of Parent-Child Activities
Description: Frequency of Parent-Child Activity measured by an additive index of survey items where number of days spent doing activity is multiplied by the number of minutes reported doing activity per day (see Appendix Table 8 in "Analysis Plan and Measures" document for items).
  Higher score indicates better outcome.
  We will estimate the statistical significance of the entire family of related measures in the Frequency of Parent-Child Activity outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Rodriguez, E. T., & Tamis-LeMonda, C. S. (2011). Trajectories of the home learning environment across the first 5 years: Associations with children's vocabulary and literacy skills at prekindergarten. Child development, 82(4), 1058-1075.
Time Frame: Age 48 months
Reporting Status: Not Posted

220. Secondary Outcome: Frequency of Parent-Child Activity: Self-Report of Parent-Child Activities
Description: Additive index of activities where the number of days reported doing the activity are multiplied by the number of minutes on a given day. We expect higher amount for high cash group. Activities are: read books, tell stories, play together, pretend play, physical games outside, learning activities, watch tv or videos. 1. How many days did you participate in [activity]? (1: no days; 2: 1-2 days; 3: 3-5 days; 4: 6-7 days) 1a. On those days, how many minutes do you do typically do this per day? (1: 15 minutes or less; 2: 15-30 minutes; 3: more than 30 minutes).
  References:
  Rodriguez, E. T., & Tamis-LeMonda, C. S. (2011). Trajectories of the home learning environment across the first 5 years: Associations with children's vocabulary and literacy skills at prekindergarten. Child development, 82(4), 1058-1075.
  BFY Study PIs
Time Frame: Age 6
Reporting Status: Not Posted

221. Secondary Outcome: Frequency of Parent-Child Activity: Self-Report of Parent-Child Activities
Description: as for outcome 220
Time Frame: Age 8
Reporting Status: Not Posted

222. Secondary Outcome: Frequency of Parent-Child Activity: Child Meal and Sleep Routine Index
Description: Frequency of Parent-Child Activity measured by an additive index of survey items (see Appendix Table 8 in "Analysis Plan and Measures" document for items).
  Minimum score: 0 Maximum score: 2. Higher score indicates better outcome.
  We will estimate the statistical significance of the entire family of related measures in the Frequency of Parent-Child Activity outcome cluster measured during the same wave using step-down resampling methods for multiple testing (see statistical analysis plan for more details; Westfall and Young, 1993).
  Reference:
  Study PIs
Time Frame: Age 48 months
Reporting Status: Not Posted

223. Secondary Outcome: Frequency of Parent-Child Activity: Child Meal and Sleep Routine Index
Description: Frequency of Parent-Child Activity measured by an additive index of survey items (see Appendix Table 10 in Statistical Analysis Plan document for items).
  Minimum score: 0 Maximum score: 2. Higher score indicates better outcome. Expect higher score for high-cash group.
  Reference:
  BFY Study PIs
Time Frame: Age 6
Reporting Status: Not Posted

224. Secondary Outcome: Frequency of Parent-Child Activity: Child Meal and Sleep Routine Index
Description: as for outcome 223
Time Frame: Age 8
Reporting Status: Not Posted

225. Secondary Outcome: Maternal Discipline: Spanking Discipline Strategy
Description: Measured by a survey item (see Appendix Table 8 in "Analysis Plan and Measures" document for items).
  Reference:
  Reichman, N.E., Teitler, J.O., Garfinkel, I., MclAnahan, S.S. (2001). Fragile Families: Sample and design. Children and Youth Services Review, 23(4-5), 303-326.
Time Frame: Age 12 months
Reporting Status: Not Posted

226. Secondary Outcome: Maternal Discipline; Spanking Discipline Strategy
Description: as for outcome 225
Time Frame: Age 24 months
Reporting Status: Not Posted

227. Secondary Outcome: Maternal Discipline; Spanking Discipline Strategy
Description: Measured by a survey item (see Appendix Table 8 in "Analysis Plan and Measures" document for items).
  Minimum score: 0; Maximum score: 1. Higher score indicates worse outcome.
  Reference:
  Reichman, N.E., Teitler, J.O., Garfinkel, I., MclAnahan, S.S. (2001). Fragile Families: Sample and design. Children and Youth Services Review, 23(4-5), 303-326.
Time Frame: Age 36 months
Reporting Status: Not Posted

228. Secondary Outcome: Maternal Discipline: Parent-Child Conflict Tactics Scale (CTSPC)
Description: Parent-Child Conflict Tactics Scale (CTSPC) Subscales: Nonviolent Discipline, Psychological Aggression, and Corporal punishment and 1 item from the Severe Assault (physical abuse) subscale. Total 14 items about conflict strategies with child and harsh discipline are asked about the past year. Min: 14 Max: 98 We expect a reduction of harsh discipline in the high-cash group compared to the low-cash group.
  References:
  Straus, M. A., Hamby, S. L., Finkelhor, D., Moore, D. W., & Runyan, D. (1998). Identification of child maltreatment with the Parent-Child Conflict Tactics Scales: Development and psychometric data for a national sample of American parents. Child abuse & neglect, 22(4), 249-270. https://doi.org/10.1016/S0145-2134(97)00174-9 Cotter, A., Proctor, K. B., & Brestan-Knight, E. (2018). Assessing child physical abuse: An examination of the factor structure and validity of the Parent-Child Conflict Tactics Scale (CTSPC). Children and Youth Services Review, 88, 467-475.
Time Frame: Age 6
Reporting Status: Not Posted

229. Secondary Outcome: Maternal Discipline: Parent-Child Conflict Tactics Scale (CTSPC)
Description: as for outcome 228
Time Frame: Age 8
Reporting Status: Not Posted

230. Secondary Outcome: Child School Retention
Description: Maternal report of whether the child has repeated a grade, adapted from the School Enrollment and Expectations section of the PSID Child Development Supplement. Item: Has child "ever" been held back a grade? Expect fewer retentions in high cash group.
  Adapted from the School Enrollment and Expectations (SEE) section of the 2021 Panel Study of Income Dynamics (PSID) Child Development Supplement: Beaule, A. Campbell, F., Insolera, N., Juska, P., McAloon-Fernandez, R., McGonagle, K., Mushtaq, M., Simmert, B., & Warra, J. (2023). PSID-2021 Main Interview User Manual: Release 2023. Institute for Social Research, University of Michigan. https://psidonline.isr.umich.edu/data/Documentation/UserGuide2021.pdf
Time Frame: Age 6
Reporting Status: Not Posted

231. Secondary Outcome: Child School Retention
Description: as for outcome 230
Time Frame: Age 8
Reporting Status: Not Posted

232. Secondary Outcome: Child Engagement in School
Description: Maternal report of child's engagement in school using an item adapted from the Survey of Income and Program Participation. "How often would you say that (CHILD) cares about doing well in school"? 4 answer choices: 1. none of the time; 2. some of the time, 3. most of the time; 4. all of the time. Score range: 1-4; higher scores indicate more engagement in school. Expect more engagement in high cash group.
  Reference: Ehrle, J. L., & Moore, K. M. (1999). 1997 NSAF Benchmarking Measures of Child and Family Well-Being. Washington, D.C.: The Urban Institute. National Survey of America's Families Methodology Report No. 6. https://webarchive.urban.org/UploadedPDF/Methodology_6.pdf
Time Frame: Age 6
Reporting Status: Not Posted

233. Secondary Outcome: Child Engagement in School
Description: as for outcome 232
Time Frame: Age 8
Reporting Status: Not Posted

234. Secondary Outcome: Child School Suspensions
Description: Maternal report of the number of school suspensions, adapted from the Survey of Income and Program Participation. One item: Has child ever been suspended or expelled from school? (no/yes). Expect fewer suspensions in high cash group.
  Reference: Adapted from the Survey of Income and Program Participation (SIPP): U.S. Census Bureau. (2023). 2022 Survey of Income and Program Participation Users' Guide. U.S. Department of Commerce Economic and Statistics Administration. https://www2.census.gov/programs-surveys/sipp/tech-documentation/methodology/2022_SIPP_Users_Guide_SEP23.pdf
Time Frame: Age 6
Reporting Status: Not Posted

235. Secondary Outcome: Child School Suspensions
Description: Maternal report of the number of school suspensions, adapted from the Survey of Income and Program Participation.One item: Has child ever been suspended or expelled from school? (no/yes). Expect fewer suspensions in high cash group.
  Reference: Adapted from the Survey of Income and Program Participation (SIPP): U.S. Census Bureau. (2023). 2022 Survey of Income and Program Participation Users' Guide. U.S. Department of Commerce Economic and Statistics Administration. https://www2.census.gov/programs-surveys/sipp/tech-documentation/methodology/2022_SIPP_Users_Guide_SEP23.pdf
Time Frame: Age 8
Reporting Status: Not Posted

236. Secondary Outcome: Child School Attendance
Description: Estimated number of days missed in last 12 months. Expect fewer absences in high-cash gift group.
  Reference: BFY Study PIs
Time Frame: Age 8
Reporting Status: Not Posted

237. Secondary Outcome: School Quality
Description: Gathered from school names and city/district. We expect an increase in school quality for the high-cash gift group. The measure we select will be a function of what data will be available at the time of Age 8 wave.
Time Frame: Age 8
Reporting Status: Not Posted

238. Secondary Outcome: Parent School Involvement
Description: Additive index of survey items (see Appendix Table 10 in Statistical Analysis Plan document for items).
  Minimum score: 0 Maximum score: 4. Higher score indicates better outcome. We expect a positive effect on high-cash group.
  Reference:
  Tourangeau, K., Nord, C., Lê, T., Wallner-Allen, K., Vaden-Kiernan, N., Blaker, L. and Najarian, M. (2019). Early Childhood Longitudinal Study, Kindergarten Class of 2010-11 (ECLS-K:2011) User's Manual for the ECLS-K:2011 Kindergarten-Fifth Grade Data File and Electronic Codebook, Public Version (NCES 2019-051). U.S. Department of Education. Washington, DC: National Center for Education Statistics. https://nces.ed.gov/pubs2019/2019051.pdf
Time Frame: Age 8
Reporting Status: Not Posted

239. Secondary Outcome: Enrichment Activities: Child Enrichment
Description: as for outcome 238
Time Frame: Age 6
Reporting Status: Not Posted

240. Secondary Outcome: Enrichment Activities: Child Enrichment
Description: as for outcome 238
Time Frame: Age 8
Reporting Status: Not Posted

241. Secondary Outcome: Enrichment Activities: Child Lessons, Sports, Etc. Activity Participation
Description: as for outcome 238
Time Frame: Age 6
Reporting Status: Not Posted

242. Secondary Outcome: Enrichment Activities: Child Lessons, Sports, Etc. Activity Participation
Description: as for outcome 238
Time Frame: Age 8
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Baseline up until our Age-4 data collection wave (i.e., 48 months).
Description: We reported the total number of mothers who died due to any cause. Note that in addition to the five mothers who died, there were five children who died due to any cause. Because our results are reported on the n=1000 mothers, we only included mothers in our reporting of adverse events.
Arm/Group | Monthly Cash Gift Payments of $333 | Monthly Cash Gift Payments of $20
All-Cause Mortality (participants affected / at risk) | 0/400 | 5/600
Serious Adverse Events (participants affected / at risk) | 0/400 | 0/600
Other Adverse Events (participants affected / at risk) | 0/400 | 0/600

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (5):
  • Study Protocol: Phase 1 Study Protocol (2019-06-27): https://cdn.clinicaltrials.gov/large-docs/56/NCT03593356/Prot_002.pdf
  • Study Protocol: Phase 2 Study Protocol (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/56/NCT03593356/Prot_011.pdf
  • Statistical Analysis Plan (2025-01-24): https://cdn.clinicaltrials.gov/large-docs/56/NCT03593356/SAP_015.pdf
  • Informed Consent Form: Age 4 Consent (2022-11-09): https://cdn.clinicaltrials.gov/large-docs/56/NCT03593356/ICF_010.pdf
  • Informed Consent Form: Age 6 Consent (2024-06-14): https://cdn.clinicaltrials.gov/large-docs/56/NCT03593356/ICF_014.pdf